CLINICAL TRIAL: NCT03784079
Title: A Randomized, Double-Blind (Sponsor-unblinded), Placebo-Controlled, Adaptive Trial to Investigate the Antiviral Effect, Safety, Tolerability and Pharmacokinetics of GSK3640254 in HIV-1 Infected Treatment-Naïve Adults
Brief Title: A Proof of Concept Study of GSK3640254 in Human Immunodeficiency Virus-1 (HIV-1) Infected Treatment-naive Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 208132
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Results first posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: HIV Infections
Keywords: HIV-1, Antiviral Effect, GSK3640254, Proof of Concept
MeSH Terms: conditions — HIV Infections | interventions — GSK3640254

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomized to receive two active doses of GSK3640254 along with placebo in Part 1 of the study. In Part 2, subjects will receive three active doses of GSK3640254 along with placebo depending upon the data obtained in Part 1.
Who Masked: Participant, Investigator
Masking Description: This will be a double blind study. Subjects and investigator will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1: GSK3640254 10 mg (Experimental): Participants will receive GSK3640254 10 milligram (mg), capsules, orally for 10 days.
  Interventions: Drug: GSK3640254
- Part 1: GSK3640254 200 mg (Experimental): Participants will receive GSK3640254 200 mg, capsules, orally for 10 days.
  Interventions: Drug: GSK3640254
- Part 1: Placebo (Placebo Comparator): Participants will receive placebo capsules, orally for 10 days.
  Interventions: Drug: Placebo matching GSK3640254 Mesylate salt
- Part 2: GSK3640254 40 mg (Experimental): Participants will receive GSK3640254 40 mg, capsules, orally for 7 days.
  Interventions: Drug: GSK3640254
- Part 2: GSK3640254 80 mg (Experimental): Participants will receive GSK3640254 80 mg, capsules, orally for 7 days.
  Interventions: Drug: GSK3640254
- Part 2: GSK3640254 140 mg (Experimental): Participants will receive GSK3640254 140 mg, capsules, orally for 7 days.
  Interventions: Drug: GSK3640254
- Part 2: Placebo (Placebo Comparator): Participants will receive placebo capsules, orally for 7 days.
  Interventions: Drug: Placebo matching GSK3640254 Mesylate salt

INTERVENTIONS:
Drug: GSK3640254 — GSK3640254 will be available with dosing strengths of 5 mg, 20 mg, and 100 mg to be administered as an oral capsule along with 240 mL of water.
  Arms: Part 1: GSK3640254 10 mg; Part 1: GSK3640254 200 mg; Part 2: GSK3640254 140 mg; Part 2: GSK3640254 40 mg; Part 2: GSK3640254 80 mg
Drug: Placebo matching GSK3640254 Mesylate salt — Placebo to match GSK3640254 Mesylate salt will be given as an oral capsule along with 240 mL of water
  Arms: Part 1: Placebo; Part 2: Placebo

SUMMARY:
Infection with HIV-1 continues to be a serious health threat throughout the world. Chronic exposure to combination anti-retroviral therapy identified anti-retroviral associated long-term toxicities. Hence, there is a need to prevent these co-morbidities. GSK3640254 is a next-generation HIV-1 Maturation Inhibitor (MI) which may be effective for HIV-1 infection. This study will evaluate the antiviral effect, safety, tolerability and pharmacokinetics/ pharmacodynamics of GSK3640254 in HIV-1 infected treatment-naive adults. This study will consists of two parts; Part 1 and Part 2. Part 1 will evaluate two active doses of GSK3640254, 200 milligrams (mg) (Cohort 1) and 10 mg (Cohort 2) along with placebo to match GSK3640254 Mesylate salt. Part 2 will evaluate three active doses of GSK3640254. Dose level 1 of GSK3640254 that can provide at least 30 percent of the maximum effect (Cohort 1), dose level 2 of GSK3640254 that can provide at least 75 percent of the maximum effect (Cohort 2) and dose level 3 of GSK3640254 that can provide at least 90 percent of the maximum effect (Cohort 3). These doses are anticipated to be 5 mg, 40 mg and 100 mg respectively, but could be modified based on data obtained in Part 1. Subjects will also receive placebo to match GSK3640254 Mesylate salt in Part 2 of the study. All doses will be administered after a moderate fat meal. This study will consist of Screening period (up to 14 days), Treatment period (Day 1- Day 10), post-dose Follow-up (Day 11- Day 17) and final Follow-up (Day 18-24). A total of approximately 34 subjects will be enrolled, of which, 14 subjects will be randomized in Part 1 and 20 in Part 2 of the study. Six subjects will be enrolled in each of the active dose cohorts and 2 subjects will be enrolled in each of the placebo cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 to 65 years of age inclusive, at the time of signing the informed consent.
* Subjects who are healthy (other than HIV infection) as determined by the Investigator or medically qualified designee based on a medical evaluation including medical history, laboratory tests, and cardiac monitoring.
* Screening Cluster of designation 4 positive (CD4+) T-cell count >=350 cells per millimeter cube (cells/mm^3).
* Documented HIV infection and Screening plasma HIV-1 RNA >=5000 copies/milliliter (mL). A single repeat of this test is allowed within a single Screening period to determine eligibility.
* Treatment-naive: No anti-retrovirals (in combination or monotherapy) received after the diagnosis of HIV-1 infection.
* Body weight >=50.0 kilograms (kg) (110 Pounds) for men and >=45.0 kg (99 pounds) for women and body mass index (BMI) within the range 18.5-31.0 kg/meter square (kg/m^2) (inclusive).
* A female subject is eligible to participate if she is not pregnant, not breastfeeding, and not a woman of childbearing potential (WOCBP).
* Capable of giving signed informed consent.
* For subjects enrolled in France: a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Presence of Hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to starting study treatment.
* Positive Hepatitis C antibody test result at screening or within 3 months prior to starting study treatment and positive on reflex to Hepatitis C RNA.
* ALT >2 times upper limit of normal (ULN). A single repeat of ALT is allowed within a single Screening period to determine eligibility.
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Subjects with primary HIV infection, evidenced by acute retroviral syndrome (example given [e.g.], fever, malaise, fatigue, etc) and/or evidence of recent (within 3 months) documented viremia without antibody production and/or evidence of recent (within 3 months) documented seroconversion.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones);
* A pre-existing condition interfering with normal gastrointestinal anatomy or motility (e.g., gastroesophageal reflux disease [GERD], gastric ulcers, gastritis), hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs or render the subject unable to take oral study treatment.
* Any acute laboratory abnormality at screen which, in the opinion of the investigator, should preclude participation in the study of an investigational compound.
* Any Grade 2-4 laboratory abnormality at screen, with the exception of creatine phosphokinase (CPK) and lipid abnormalities (e.g., total cholesterol, triglycerides, etc), and ALT (described above), will exclude a subject from the study unless the investigator can provide a compelling explanation for the laboratory result(s) and has the assent of the sponsor. A single repeat of any lab abnormality is allowed within a single screening period to determine eligibility.
* Any history of significant underlying psychiatric disorder, including but not limited to schizophrenia, bipolar disorder with or without psychotic symptoms, other psychotic disorders, or schizotypal (personality) disorder.
* Any history of major depressive disorder with or without suicidal features, or anxiety disorders, that required medical intervention (pharmacologic or not) such as hospitalization or other inpatient treatment and/or chronic (>6 months) outpatient treatment. Subjects with other conditions such as adjustment disorder or dysthymia that have required shorter term medical therapy (<6 months) without inpatient treatment and are currently well-controlled clinically or resolved may be considered for entry after discussion and agreement with the ViiV Medical Monitor.
* Any pre-existing physical or other psychiatric condition (including alcohol or drug abuse), which, in the opinion of the investigator (with or without psychiatric evaluation), could interfere with the subject's ability to comply with the dosing schedule and protocol evaluations or which might compromise the safety of the subject.
* Medical history of cardiac arrhythmias or cardiac disease or a family or personal history of long QT syndrome.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* The subject has participated in a clinical trial and has received an investigational product within the 30 days prior to the first dosing day in the current study.
* Any positive (abnormal) response confirmed by the investigator on a Screening clinician- (or qualified designee-) administered Columbia Suicide Severity Rating Scale (CSSRS).
* Any positive result for illicit drug use (e.g., cocaine, heroin) at Screening. A positive screen for marijuana is not exclusionary, though if positive for delta-9-tetrahydrocannabinol (THC).
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56 days.
* Exposure to more than four new investigational drugs or vaccines within 12 months prior to the first dosing day.
* Treatment with radiation therapy or cytotoxic chemotherapeutic agents within 30 days of study drug administration or anticipated need for such treatment within the study.
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical, anal or penile intraepithelial neoplasia; or other localized malignancies require agreement between the investigator and the study medical monitor for inclusion of the subject prior to randomization.
* Treatment with immunomodulating agents (such as systemic corticosteroids, interleukins, interferons) or any agent with known anti-HIV activity (such as hydroxyurea or foscarnet) within 30 days of study drug administration.
* An active Center for Disease Control and Prevention (CDC) Category C disease except cutaneous Kaposi's sarcoma not requiring systemic therapy during the trial.
* Treatment with any vaccine within 30 days prior to receiving study medication.
* Exclusion criteria for screening electrocardiogram (a single repeat is allowed for eligibility determination): Heart rate of <45 or >100 beats per minute (bpm) for males and <50 or >100 bpm for females; PR Interval of <120 or >200 milliseconds (msec) for both males and females; QRS duration of <70 or >110 msec for both males and females; QT interval corrected (QTc) for heart rate according to Fridericia's formula (QTcF) of >450 msec for males and >470 msec for females. A heart rate from 100 to 110 bpm can be rechecked by electrocardiogram or vitals within 30 minutes to verify eligibility. QTcF is either machine read or manually over-read.
* Any significant arrhythmia or electrocardiogram finding (e.g., prior myocardial infarction, sinoatrial pauses, bundle branch block, or conduction abnormality) which, in the opinion of the Investigator OR ViiV Medical Monitor, will interfere with the safety for the individual subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (17):
- United States (2):
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Orlando, Florida
- France (3):
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Tourcoing
- Germany (2):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
- Italy (2):
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
- South Africa (3):
  - GSK Investigational Site, Johannesburg, Gauteng
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Durban
- Spain (5):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Spinner CD, Felizarta F, Rizzardini G, Philibert P, Mitha E, Domingo P, Stephan CJ, DeGrosky M, Bainbridge V, Zhan J, Dumitrescu TP, Jeffrey JL, Xu J, Halliday F, Gan J, Johnson M, Gartland M, Joshi SR, Lataillade M. Phase IIa Proof-of-Concept Evaluation of the Antiviral Efficacy, Safety, Tolerability, and Pharmacokinetics of the Next-Generation Maturation Inhibitor GSK3640254. Clin Infect Dis. 2022 Sep 14;75(5):786-794. doi: 10.1093/cid/ciab1065. PMID 34996113

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, double-blind, placebo-controlled, adaptive clinical trial to evaluate the antiviral effect, safety, tolerability and pharmacokinetic (PK)/pharmacodynamics (PD) of GSK3640254 over 10 days in study Part 1 and over 7 days in study Part 2.
Pre-assignment Details: A total of 34 participants (14 participants in Part 1 and 20 participants in Part 2) were enrolled in this study. This study was conducted in France, Germany, Italy, South Africa and Spain.
Groups:
- Part 1: GSK3640254 10 mg: Participants received GSK3640254 10 milligram (mg), capsules, orally for 10 days. Participants were followed for up to 14 days post last dose of study treatment.
- Part 1: GSK3640254 200 mg: Participants received GSK3640254 200 mg, capsules, orally for 10 days. Participants were followed for up to 14 days post last dose of study treatment.
- Part 1: Placebo: Participants received placebo capsules, orally for 10 days. Participants were followed for up to 14 days post last dose of study treatment.
- Part 2: GSK3640254 40 mg: Participants received GSK3640254 40 mg, capsules, orally for 7 days. Participants were followed for up to 5 days post last dose of study treatment.
- Part 2: GSK3640254 80 mg: Participants received GSK3640254 80 mg, capsules, orally for 7 days. Participants were followed for up to 5 days post last dose of study treatment.
- Part 2: GSK3640254 140 mg: Participants received GSK3640254 140 mg, capsules, orally for 7 days. Participants were followed for up to 5 days post last dose of study treatment.
- Part 2: Placebo: Participants received placebo capsules, orally for 7 days. Participants were followed for up to 5 days post last dose of study treatment.
Period: Part 1: Up to Day 24
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Started | 6 | 6 | 2 | 0 | 0 | 0 | 0
Completed | 6 | 6 | 2 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Up to Day 12
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Started | 0 | 0 | 0 | 6 | 6 | 6 | 2
Completed | 0 | 0 | 0 | 6 | 6 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1: GSK3640254 10 mg: Participants received GSK3640254 10 mg, capsules, orally for 10 days. Participants were followed for up to 14 days post last dose of study treatment.
- Total: Total of all reporting groups
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo | Total
Number analyzed (Participants) | 6 | 6 | 2 | 6 | 6 | 6 | 2 | 34
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  19-64 years | 6 | 6 | 2 | 6 | 6 | 6 | 2 | 34
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Male | 6 | 6 | 2 | 5 | 6 | 5 | 2 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  Asian: South East Asian Heritage | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 4
  White: White/Caucasian/European Heritage | 2 | 5 | 2 | 5 | 4 | 5 | 1 | 24
  Multiple: American Indian or Alaska Native & White | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Maximum Change From Baseline in Plasma Human Immunodeficiency Virus-1 (HIV-1) Ribonucleic Acid (RNA) at Day 11
Description: Plasma samples were collected for quantitative analysis of plasma HIV-1 RNA. A HIV-1 RNA polymerase chain reaction (PCR) assay with a lower limit of detection (LLOD) of 50 copies per milliliter was used. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Day 11
Population: Intent-To-Treat Exposed Population consisted of all participants who met study criteria and were enrolled into the study with documented evidence of having received at least 1 dose of treatment and at least one post-Baseline HIV-1 RNA measurement.
Measure: Mean (Standard Deviation); unit: Copies per milliliter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Copies per milliliter | -8605.8 (4604.40) | -100719.8 (89182.99) | -3406.5 (2591.55)

2. Primary Outcome: Part 2: Maximum Change From Baseline in Plasma HIV-1 RNA at Day 8
Description: Plasma samples were collected for quantitative analysis of plasma HIV-1 RNA. An HIV-1 RNA PCR assay with an LLOD of 50 copies per milliliter was used. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Day 8
Population: Intent-To-Treat Exposed Population.
Measure: Mean (Standard Deviation); unit: Copies per milliliter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Copies per milliliter | -48655.0 (26269.41) | -37904.3 (38814.54) | -64904.2 (83798.67) | -123478.5 (175276.92)

3. Secondary Outcome: Part 1: Number of Participants With Non-Serious Adverse Events (Non-SAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or other situations as per Medical or scientific judgment. Safety Population consisted of all participants who were enrolled into the study with documented evidence of having received at least 1 dose of randomized treatment.
Time Frame: Up to Day 24
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Participants
  Non-SAEs | 3 | 5 | 0
  SAEs | 1 | 0 | 0

4. Secondary Outcome: Part 2: Number of Participants With Non-SAEs and SAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or other situations as per Medical or scientific judgment.
Time Frame: Up to Day 12
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Participants
  Non-SAEs | 5 | 4 | 4 | 0
  SAEs | 0 | 0 | 1 | 0

5. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Leukocytes, Platelet Count
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the hematology parameters: basophils, eosinophils, lymphocytes, monocytes, neutrophils, leukocytes and platelet count. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
10^9 cells per liter
  Basophils | 0.005 (0.0266) | -0.017 (0.0234) | 0.015 (0.0212)
  Eosinophils | -0.023 (0.1296) | 0.058 (0.1134) | -0.025 (0.0212)
  Lymphocytes | -0.027 (0.5267) | 0.458 (0.4412) | 0.070 (0.0566)
  Monocytes | 0.100 (0.1124) | -0.000 (0.0980) | 0.055 (0.0212)
  Neutrophils | -0.045 (0.4624) | -0.525 (0.8169) | 0.345 (0.1485)
  Leukocytes | 0.02 (0.679) | -0.02 (1.057) | 0.45 (0.212)
  Platelet count | 25.0 (46.35) | 11.8 (12.04) | 13.0 (2.83)

6. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the hematology parameter: hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Grams per liter | -4.2 (4.96) | -1.8 (5.98) | -1.0 (5.66)

7. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the hematology parameter: hematocrit. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Proportion of red blood cells in blood | -0.0117 (0.01684) | -0.0073 (0.01919) | -0.0010 (0.01838)

8. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameter: Erythrocytes
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the hematology parameter: erythrocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
10^12 cells per liter | -0.10 (0.190) | -0.07 (0.197) | 0.00 (0.141)

9. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the hematology parameter: erythrocytes mean corpuscular volume. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Femtoliter | 0.0 (0.89) | -0.3 (1.03) | 0.0 (0.00)

10. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Picograms | -0.08 (0.286) | 0.03 (0.266) | -0.15 (0.071)

11. Secondary Outcome: Part 1: Change From Baseline in Hematology Parameter: Reticulocytes/Erythrocyte
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the hematology parameter: reticulocytes/erythrocyte (erythro). Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Percentage of reticulocytes in erythro
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Percentage of reticulocytes in erythro | 0.0042 (0.00449) | 0.0012 (0.00172) | 0.0020 (0.00000)

12. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Leukocytes, Platelet Count
Description: Blood samples were collected to analyze the hematology parameters: basophils, eosinophils, lymphocytes, monocytes, neutrophils, leukocytes and platelet count. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles).
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 2
10^9 cells per liter
  Basophils, n=5,6,5,2: number analyzed (Participants) | 5 | 6 | 5 | 2
  Basophils, n=5,6,5,2 | 0.010 (0.0141) | 0.020 (0.0237) | 0.022 (0.0084) | -0.005 (0.0354)
  Eosinophils, n=5,6,5,2: number analyzed (Participants) | 5 | 6 | 5 | 2
  Eosinophils, n=5,6,5,2 | -0.066 (0.2145) | -0.047 (0.1775) | 0.034 (0.0404) | 0.020 (0.0000)
  Lymphocytes, n=5,6,5,2: number analyzed (Participants) | 5 | 6 | 5 | 2
  Lymphocytes, n=5,6,5,2 | 0.006 (0.4458) | -0.062 (0.4731) | 0.536 (0.4766) | -0.110 (0.2687)
  Monocytes, n=5,6,5,2: number analyzed (Participants) | 5 | 6 | 5 | 2
  Monocytes, n=5,6,5,2 | -0.020 (0.0869) | 0.022 (0.1705) | -0.084 (0.1436) | -0.130 (0.1131)
  Neutrophils, n=5,6,5,2: number analyzed (Participants) | 5 | 6 | 5 | 2
  Neutrophils, n=5,6,5,2 | 0.424 (0.6401) | 1.678 (2.1754) | 0.432 (0.7007) | -0.215 (0.3182)
  Leukocytes, n=5,6,6,2 | 0.34 (0.385) | 1.62 (2.244) | 0.52 (1.211) | -0.45 (0.071)
  Platelet count, n=4,6,6,2: number analyzed (Participants) | 4 | 6 | 6 | 2
  Platelet count, n=4,6,6,2 | 1.5 (45.82) | 17.5 (30.26) | 16.0 (21.57) | 4.5 (0.71)

13. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 2
Grams per liter | -8.0 (5.10) | -4.7 (6.59) | -1.7 (7.31) | -8.0 (1.41)

14. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 2
Proportion of red blood cells in blood | -0.0230 (0.01762) | -0.0123 (0.02096) | -0.0058 (0.02094) | -0.0315 (0.01485)

15. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 2
10^12 cells per liter | -0.24 (0.207) | -0.17 (0.216) | -0.08 (0.223) | -0.30 (0.000)

16. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular volume. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 2
Femtoliter | -0.2 (0.45) | 0.2 (0.98) | 0.2 (0.98) | -2.0 (2.83)

17. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 2
Picograms | -0.28 (0.850) | -0.05 (0.187) | -0.02 (0.337) | -0.05 (0.354)

18. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Reticulocytes/Erythro
Description: Blood samples were collected to analyze the hematology parameter: reticulocytes/erythro. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of reticulocytes in erythro
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 2
Percentage of reticulocytes in erythro | 0.0030 (0.00235) | 0.0017 (0.00258) | 0.0007 (0.00350) | 0.0020 (0.00283)

19. Secondary Outcome: Part 1: Change From Baseline in Chemistry Parameters: Glucose, Cholesterol, Triglycerides, Calcium, Chloride, Phosphate, Potassium, Magnesium, Sodium, Urea, High Density Lipoprotein (HDL) Cholesterol, Low Density Lipoprotein (LDL) Cholesterol
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the chemistry parameters: glucose, cholesterol, triglycerides, calcium, chloride, phosphate, potassium, magnesium, sodium, urea, HDL cholesterol and LDL cholesterol. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Millimoles per liter
  Glucose, n=6,6,2 | -0.20 (0.253) | 0.28 (0.595) | 0.00 (0.424)
  Cholesterol, n=0,0,0: number analyzed (Participants) | 0 | 0 | 0
  Triglycerides, n=0,0,0: number analyzed (Participants) | 0 | 0 | 0
  Calcium, n=6,6,2 | -0.007 (0.1343) | -0.027 (0.0468) | 0.020 (0.0283)
  Chloride, n=6,6,2 | 0.0 (2.10) | 0.8 (3.06) | -0.5 (3.54)
  Phosphate, n=6,6,2 | 0.042 (0.1594) | 0.058 (0.1772) | -0.075 (0.1061)
  Potassium, n=6,6,2 | 0.02 (0.240) | -0.03 (0.242) | -0.10 (0.000)
  Magnesium, n=6,6,2 | 0.000 (0.0551) | -0.007 (0.0561) | -0.020 (0.0283)
  Sodium, n=6,6,2 | 0.2 (2.40) | -0.8 (1.60) | -1.0 (1.41)
  Urea, n=6,6,2 | -0.08 (1.021) | -0.08 (0.801) | 1.00 (0.000)
  HDL cholesterol, n=0,0,0: number analyzed (Participants) | 0 | 0 | 0
  LDL cholesterol, n=0,0,0: number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: Part 1: Change From Baseline in Chemistry Parameters: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST)
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the chemistry parameters: ALT, ALP and AST. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
International units per liter
  ALT | 2.7 (7.79) | -1.7 (4.46) | 9.5 (6.36)
  ALP | 10.5 (23.36) | -3.5 (4.64) | -4.0 (1.41)
  AST | -0.5 (3.94) | -2.0 (8.60) | 4.5 (2.12)

21. Secondary Outcome: Part 1: Change From Baseline in Chemistry Parameters: Creatinine, Bilirubin
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the chemistry parameters: creatinine and bilirubin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Micromoles per liter
  Creatinine | 1.77 (5.565) | -1.33 (4.291) | 0.00 (0.000)
  Bilirubin | -0.3 (3.20) | -2.0 (2.53) | 3.0 (9.90)

22. Secondary Outcome: Part 1: Change From Baseline in Chemistry Parameters: Protein
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the chemistry parameter: protein. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Grams per liter | -1.3 (4.93) | -1.0 (2.97) | 1.0 (2.83)

23. Secondary Outcome: Part 1: Change From Baseline in Chemistry Parameters: Amylase, Lipase
Description: Blood samples were collected to analyze the chemistry parameters: amylase and lipase. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 6 (Day 11)
Population: Safety Population. Only those participants with data available at the specified time points were analyzed. Amylase and lipase results were collected for two participants in GSK3640254 10 mg arm during Part 1 of the study. No data were collected for Placebo and GSK3640254 200 mg arms at Visit 6 (Day 11) due to delays in approval of Protocol Amendment 02 into which testing for amylase and lipase was added.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 2 | 0 | 0
Units per liter
  Amylase | 0.0 (11.31) |  |
  Lipase | -2.0 (2.83) |  |

24. Secondary Outcome: Part 2: Change From Baseline in Chemistry Parameters: Glucose, Cholesterol, Triglycerides, Calcium, Chloride, Phosphate, Potassium, Magnesium, Sodium, Urea, HDL Cholesterol, LDL Cholesterol
Description: Blood samples were collected to analyze the chemistry parameters: glucose, cholesterol, triglycerides, calcium, chloride, phosphate, potassium, magnesium, sodium, urea, HDL cholesterol and LDL cholesterol. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 1
Millimoles per liter
  Glucose, n=6,6,6,1 | -0.05 (0.327) | 0.18 (1.085) | -0.03 (0.446) | 0.50 (NA) — Standard deviation could not be calculated for single participant.
  Cholesterol, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Triglycerides, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Calcium, n=6,6,6,1 | -0.057 (0.0638) | -0.027 (0.0628) | 0.030 (0.1002) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Chloride, n=6,6,6,1 | -0.7 (2.25) | -0.2 (1.47) | -0.7 (2.34) | -2.0 (NA) — Standard deviation could not be calculated for single participant.
  Phosphate, n=6,6,6,1 | -0.117 (0.2160) | 0.067 (0.1211) | 0.083 (0.1329) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Potassium, n=6,6,6,1 | -0.20 (0.261) | 0.05 (0.383) | 0.20 (0.210) | -0.10 (NA) — Standard deviation could not be calculated for single participant.
  Magnesium, n=6,6,6,1 | 0.007 (0.0484) | 0.007 (0.0413) | 0.027 (0.0501) | 0.000 (NA) — Standard deviation could not be calculated for single participant.
  Sodium, n=6,6,6,1 | -0.8 (2.23) | -0.3 (1.37) | -0.2 (1.72) | -4.0 (NA) — Standard deviation could not be calculated for single participant.
  Urea, n=6,6,6,1 | -0.42 (0.861) | -0.25 (1.037) | -0.33 (0.931) | -0.50 (NA) — Standard deviation could not be calculated for single participant.
  HDL cholesterol, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  LDL cholesterol, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0

25. Secondary Outcome: Part 2: Change From Baseline in Chemistry Parameters: ALT, ALP, AST
Description: Blood samples were collected to analyze the chemistry parameters: ALT, ALP and AST. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 1
International units per liter
  ALT | -3.8 (6.62) | -1.2 (3.76) | -6.2 (8.33) | -1.0 (NA) — Standard deviation could not be calculated for single participant.
  ALP | -3.2 (3.19) | -0.7 (5.35) | -1.8 (8.61) | -1.0 (NA) — Standard deviation could not be calculated for single participant.
  AST | -5.2 (9.37) | 0.3 (5.79) | -4.7 (7.37) | 4.0 (NA) — Standard deviation could not be calculated for single participant.

26. Secondary Outcome: Part 2: Change From Baseline in Chemistry Parameters: Creatinine, Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: creatinine and bilirubin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 1
Micromoles per liter
  Creatinine | 1.35 (3.230) | -3.38 (2.230) | -0.17 (8.362) | -0.90 (NA) — Standard deviation could not be calculated for single participant.
  Bilirubin | -0.3 (2.34) | 1.3 (6.02) | 0.3 (1.51) | 0.0 (NA) — Standard deviation could not be calculated for single participant.

27. Secondary Outcome: Part 2: Change From Baseline in Chemistry Parameters: Protein
Description: Blood samples were collected to analyze the chemistry parameter: protein. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 1
Grams per liter | -2.2 (3.25) | -0.8 (4.07) | 1.5 (4.64) | -2.0 (NA) — Standard deviation could not be calculated for single participant.

28. Secondary Outcome: Part 2: Change From Baseline in Chemistry Parameters: Amylase, Lipase
Description: as for outcome 23
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 1
Units per liter
  Amylase | -2.3 (8.62) | 0.8 (9.87) | 6.7 (7.84) | -10.0 (NA) — Standard deviation could not be calculated for single participant.
  Lipase | -1.0 (8.27) | -2.2 (6.37) | 4.5 (8.29) | 8.0 (NA) — Standard deviation could not be calculated for single participant.

29. Secondary Outcome: Part 1: Change From Baseline in Urinalysis Parameter: Specific Gravity
Description: Urine samples were collected at Baseline and one sample between Days 8 to 10 to analyze the urinalysis parameter: specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Ratio | 0.0002 (0.00615) | 0.0008 (0.00232) | 0.0000 (0.00283)

30. Secondary Outcome: Part 1: Change From Baseline in Urinalysis Parameter: Urobilinogen
Description: Urine samples were collected at Baseline and one sample between Days 8 to 10 to analyze the urinalysis parameter: urobilinogen. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Micromoles per liter | 4.50 (6.971) | 0.00 (0.000) | 0.00 (0.000)

31. Secondary Outcome: Part 1: Change From Baseline in Urinalysis Parameter: Potential of Hydrogen (pH)
Description: Urine samples were collected at Baseline and one sample between Days 8 to 10 to analyze the urinalysis parameter: pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acidic pH (5.0 - 6.0). Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
pH | 0.17 (1.033) | -0.33 (0.683) | -0.50 (0.000)

32. Secondary Outcome: Part 2: Change From Baseline in Urinalysis Parameter: Specific Gravity
Description: Urine samples were collected to analyze the urinalysis parameter: specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Ratio | 0.0010 (0.00746) | -0.0022 (0.00794) | 0.0018 (0.00744) | -0.0110 (0.00424)

33. Secondary Outcome: Part 2: Change From Baseline in Urinalysis Parameter: Urobilinogen
Description: Urine samples were collected to analyze the urinalysis parameter: urobilinogen. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Micromoles per liter | 0.00 (0.000) | 4.50 (6.971) | 0.00 (0.000) | 0.00 (0.000)

34. Secondary Outcome: Part 2: Change From Baseline in Urinalysis Parameter: pH
Description: Urine samples were collected to analyze the urinalysis parameter: pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acidic pH (5.0 - 6.0). Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
pH | 0.17 (0.683) | -0.17 (0.683) | 0.08 (0.492) | 0.25 (0.354)

35. Secondary Outcome: Part 1: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured in the semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Millimeters of mercury
  SBP | -2.5 (8.41) | 0.5 (9.65) | -1.5 (3.54)
  DBP | -0.3 (14.50) | 0.8 (4.67) | 0.5 (0.71)

36. Secondary Outcome: Part 1: Change From Baseline in Respiratory Rate
Description: Respiratory rate was measured in the semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Breaths per minute | -1.0 (1.79) | 0.2 (2.32) | -1.0 (1.41)

37. Secondary Outcome: Part 1: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in the semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Beats per minute | -5.2 (4.36) | 5.5 (10.99) | 6.0 (2.83)

38. Secondary Outcome: Part 2: Change From Baseline in SBP and DBP
Description: as for outcome 35
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Millimeters of mercury
  SBP | 1.0 (8.27) | -2.2 (4.45) | 7.3 (11.55) | 1.0 (2.83)
  DBP | -1.8 (2.40) | -1.0 (6.36) | 2.3 (15.72) | -0.5 (7.78)

39. Secondary Outcome: Part 2: Change From Baseline in Respiratory Rate
Description: as for outcome 36
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Breaths per minute | -0.2 (1.83) | 0.2 (1.47) | -1.0 (4.47) | 0.5 (2.12)

40. Secondary Outcome: Part 2: Change From Baseline in Pulse Rate
Description: as for outcome 37
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Beats per minute | 4.2 (17.36) | 2.0 (11.14) | 2.8 (6.40) | 10.5 (7.78)

41. Secondary Outcome: Part 1: Change From Baseline in Electrocardiogram (ECG) Parameters: PR Interval, QRS Duration, QT Interval, Corrected QT Interval Using Bazett's Formula (QTcB), Corrected QT Interval Using Fridericia's Formula (QTcF)
Description: Twelve lead ECGs were obtained to measure PR Interval, QRS Duration, QT Interval, QTcB Interval and QTcF Interval. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value.
Time Frame: Baseline (Day 1), Visit 5 (Days 8 to 10: Pre-dose, 2, 4 and 6 hours)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Milliseconds
  PR Interval- Days 8 to 10: Pre-dose | -0.4 (5.32) | -7.6 (5.69) | -2.5 (2.12)
  PR Interval- Days 8 to 10: 2 hours | 1.4 (5.47) | -6.3 (9.71) | -11.5 (0.71)
  PR Interval- Days 8 to 10: 4 hours | -0.1 (10.00) | 0.2 (9.81) | -3.5 (0.71)
  PR Interval- Days 8 to 10: 6 hours | 1.4 (13.22) | -5.9 (3.93) | -25.0 (4.24)
  QRS Duration- Days 8 to 10: Pre-dose | -3.1 (6.65) | -3.4 (9.90) | -5.3 (3.30)
  QRS Duration- Days 8 to 10: 2 hours | -2.1 (6.60) | 0.4 (6.27) | 0.2 (4.01)
  QRS Duration- Days 8 to 10: 4 hours | -3.3 (3.50) | -1.7 (6.75) | -1.3 (3.77)
  QRS Duration- Days 8 to 10: 6 hours | -3.6 (5.56) | -2.9 (4.55) | -2.3 (13.20)
  QT Interval- Days 8 to 10: Pre-dose | 0.7 (8.15) | -2.7 (19.60) | -19.7 (21.21)
  QT Interval- Days 8 to 10: 2 hours | -2.4 (17.61) | 4.4 (20.33) | -28.7 (4.24)
  QT Interval- Days 8 to 10: 4 hours | 8.7 (18.43) | 8.9 (13.72) | -25.2 (19.09)
  QT Interval- Days 8 to 10: 6 hours | 5.7 (16.48) | 5.8 (14.19) | -24.2 (21.92)
  QTcB Interval- Days 8 to 10: Pre-dose | 1.65 (15.813) | 3.60 (18.218) | -1.38 (6.435)
  QTcB Interval- Days 8 to 10: 2 hours | -10.45 (22.433) | -4.60 (14.266) | -27.38 (32.315)
  QTcB Interval- Days 8 to 10: 4 hours | 0.77 (15.517) | -10.37 (20.176) | -30.23 (51.760)
  QTcB Interval- Days 8 to 10: 6 hours | 2.65 (13.391) | -9.15 (15.513) | -4.88 (11.102)
  QTcF Interval- Days 8 to 10: Pre-dose | 1.2 (10.75) | 1.2 (9.56) | -7.7 (11.31)
  QTcF Interval- Days 8 to 10: 2 hours | -7.5 (19.44) | -1.3 (14.06) | -27.7 (22.63)
  QTcF Interval- Days 8 to 10: 4 hours | 3.7 (15.18) | -3.7 (10.84) | -28.7 (41.01)
  QTcF Interval- Days 8 to 10: 6 hours | 4.0 (12.82) | -3.8 (13.06) | -12.2 (14.85)

42. Secondary Outcome: Part 2: Change From Baseline in ECG Parameters: PR Interval, QRS Duration, QT Interval, QTcB, QTcF
Description: as for outcome 41
Time Frame: Baseline (Day 1), Visit 5 (Day 7: Pre-dose, 2, 4 and 6 hours)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Milliseconds
  PR Interval- Day 7: Pre-dose | 9.7 (13.92) | -1.1 (6.89) | -7.3 (9.20) | -7.3 (0.47)
  PR Interval- Day 7: 2 hours | 6.1 (14.20) | -2.4 (7.90) | -3.1 (8.61) | 6.2 (2.59)
  PR Interval- Day 7: 4 hours | 5.2 (22.87) | 1.1 (8.56) | -8.3 (6.81) | 4.7 (5.19)
  PR Interval- Day 7: 6 hours | 3.9 (16.80) | -2.3 (6.24) | -2.1 (5.82) | -7.8 (9.66)
  QRS Duration- Day 7: Pre-dose | 3.9 (5.11) | 3.2 (7.81) | -0.4 (6.87) | 2.3 (7.07)
  QRS Duration- Day 7: 2 hours | 2.4 (4.18) | 0.7 (4.89) | -0.1 (8.45) | 4.3 (1.41)
  QRS Duration- Day 7: 4 hours | 1.7 (4.06) | 0.1 (4.41) | -3.1 (6.25) | 3.8 (3.54)
  QRS Duration- Day 7: 6 hours | 0.5 (11.78) | -0.1 (3.04) | -0.8 (3.70) | 2.8 (6.36)
  QT Interval- Day 7: Pre-dose | -7.4 (33.78) | -1.6 (13.03) | 5.0 (20.49) | 3.2 (2.59)
  QT Interval- Day 7: 2 hours | -24.4 (33.17) | -4.4 (8.90) | 1.8 (12.60) | -0.3 (6.13)
  QT Interval- Day 7: 4 hours | -12.8 (25.96) | 4.2 (12.84) | -1.7 (13.65) | 11.2 (19.56)
  QT Interval- Day 7: 6 hours | -21.4 (36.18) | 5.9 (12.19) | 0.7 (12.92) | 2.7 (7.54)
  QTcB Interval- Day 7: Pre-dose | -4.16 (14.780) | 0.34 (11.468) | 3.45 (6.785) | -7.08 (2.569)
  QTcB Interval- Day 7: 2 hours | 2.90 (19.936) | 0.09 (14.494) | -4.88 (17.444) | -18.23 (2.923)
  QTcB Interval- Day 7: 4 hours | -6.96 (23.150) | -0.56 (13.559) | 1.30 (14.341) | -23.83 (2.781)
  QTcB Interval- Day 7: 6 hours | -3.26 (16.691) | 4.17 (12.302) | -1.68 (10.181) | -9.83 (17.489)
  QTcF Interval- Day 7: Pre-dose | -5.9 (18.89) | -0.5 (4.12) | 4.1 (9.23) | -3.3 (0.94)
  QTcF Interval- Day 7: 2 hours | -7.2 (22.91) | -1.3 (8.73) | -2.3 (12.87) | -12.3 (0.47)
  QTcF Interval- Day 7: 4 hours | -9.4 (21.24) | 1.2 (8.15) | 0.6 (9.00) | -12.3 (4.71)
  QTcF Interval- Day 7: 6 hours | -9.5 (19.08) | 4.5 (5.69) | -0.8 (7.79) | -5.8 (8.72)

43. Secondary Outcome: Part 1: Absolute Values for Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Leukocytes, Platelet Count
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the hematology parameters: basophils, eosinophils, lymphocytes, monocytes, neutrophils, leukocytes and platelet count. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
10^9 cells per liter
  Baseline (Day 1): Basophils, n=6,5,2: number analyzed (Participants) | 6 | 5 | 2
  Baseline (Day 1): Basophils, n=6,5,2 | 0.052 (0.0279) | 0.056 (0.0321) | 0.030 (0.0000)
  Days 8 to 10: Basophils, n=6,6,2 | 0.057 (0.0266) | 0.037 (0.0186) | 0.045 (0.0212)
  Baseline (Day 1): Eosinophils, n=6,5,2: number analyzed (Participants) | 6 | 5 | 2
  Baseline (Day 1): Eosinophils, n=6,5,2 | 0.212 (0.1783) | 0.150 (0.0616) | 0.105 (0.0212)
  Days 8 to 10: Eosinophils, n=6,6,2 | 0.188 (0.0873) | 0.202 (0.1003) | 0.080 (0.0424)
  Baseline (Day 1): Lymphocytes, n=6,5,2: number analyzed (Participants) | 6 | 5 | 2
  Baseline (Day 1): Lymphocytes, n=6,5,2 | 2.303 (0.5431) | 1.810 (0.4341) | 2.010 (0.0707)
  Days 8 to 10: Lymphocytes, n=6,6,2 | 2.277 (0.4484) | 2.217 (0.6693) | 2.080 (0.1273)
  Baseline (Day 1): Monocytes, n=6,5,2: number analyzed (Participants) | 6 | 5 | 2
  Baseline (Day 1): Monocytes, n=6,5,2 | 0.552 (0.2033) | 0.530 (0.1814) | 0.460 (0.0000)
  Days 8 to 10: Monocytes, n=6,6,2 | 0.652 (0.1907) | 0.508 (0.2088) | 0.515 (0.0212)
  Baseline (Day 1): Neutrophils, n=6,5,2: number analyzed (Participants) | 6 | 5 | 2
  Baseline (Day 1): Neutrophils, n=6,5,2 | 2.935 (0.4803) | 3.094 (0.7279) | 1.840 (0.4101)
  Days 8 to 10: Neutrophils, n=6,6,2 | 2.890 (0.6049) | 2.635 (0.4068) | 2.185 (0.2616)
  Baseline (Day 1): Leukocytes, n=6,5,2: number analyzed (Participants) | 6 | 5 | 2
  Baseline (Day 1): Leukocytes, n=6,5,2 | 6.05 (1.071) | 5.64 (1.172) | 4.45 (0.495)
  Days 8 to 10: Leukocytes, n=6,6,2 | 6.07 (0.929) | 5.60 (1.158) | 4.90 (0.283)
  Baseline (Day 1): Platelet count, n=6,5,2: number analyzed (Participants) | 6 | 5 | 2
  Baseline (Day 1): Platelet count, n=6,5,2 | 208.8 (38.48) | 202.0 (39.26) | 195.5 (12.02)
  Days 8 to 10: Platelet count, n=6,6,2 | 233.8 (70.34) | 205.0 (43.38) | 208.5 (14.85)

44. Secondary Outcome: Part 1: Absolute Values for Hematology Parameter: Hemoglobin
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the hematology parameter: hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Grams per liter
  Baseline (Day 1): n=6,5,2: number analyzed (Participants) | 6 | 5 | 2
  Baseline (Day 1): n=6,5,2 | 144.2 (11.55) | 135.4 (9.42) | 148.0 (4.24)
  Days 8 to 10: n=6,6,2 | 140.0 (12.18) | 138.7 (12.72) | 147.0 (9.90)

45. Secondary Outcome: Part 1: Absolute Values for Hematology Parameter: Hematocrit
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the hematology parameter: hematocrit. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Proportion of red blood cells in blood
  Baseline (Day 1): n=6,5,2: number analyzed (Participants) | 6 | 5 | 2
  Baseline (Day 1): n=6,5,2 | 0.4338 (0.02709) | 0.4112 (0.02523) | 0.4395 (0.01344)
  Days 8 to 10: n=6,6,2 | 0.4222 (0.03456) | 0.4158 (0.02827) | 0.4385 (0.03182)

46. Secondary Outcome: Part 1: Absolute Values for Hematology Parameter: Erythrocytes
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the hematology parameter: erythrocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
10^12 cells per liter
  Baseline (Day 1): n=6,5,2: number analyzed (Participants) | 6 | 5 | 2
  Baseline (Day 1): n=6,5,2 | 4.90 (0.228) | 4.58 (0.259) | 4.90 (0.283)
  Days 8 to 10: n=6,6,2 | 4.80 (0.290) | 4.63 (0.327) | 4.90 (0.424)

47. Secondary Outcome: Part 1: Absolute Values for Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the hematology parameter: erythrocytes mean corpuscular volume. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Femtoliter
  Baseline (Day 1): n=6,5,2: number analyzed (Participants) | 6 | 5 | 2
  Baseline (Day 1): n=6,5,2 | 88.5 (3.67) | 90.2 (3.49) | 90.0 (1.41)
  Days 8 to 10: n=6,6,2 | 88.5 (4.09) | 90.0 (2.28) | 90.0 (1.41)

48. Secondary Outcome: Part 1: Absolute Values for Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Picograms
  Baseline (Day 1): n=6,5,2: number analyzed (Participants) | 6 | 5 | 2
  Baseline (Day 1): n=6,5,2 | 29.38 (1.780) | 29.64 (0.879) | 30.25 (0.636)
  Days 8 to 10: n=6,6,2 | 29.30 (1.747) | 29.97 (0.942) | 30.10 (0.707)

49. Secondary Outcome: Part 1: Absolute Values for Hematology Parameter: Reticulocytes/Erythro
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the hematology parameter: reticulocytes/erythro. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percentage of reticulocytes in erythro
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Percentage of reticulocytes in erythro
  Baseline (Day 1): n=6,5,2: number analyzed (Participants) | 6 | 5 | 2
  Baseline (Day 1): n=6,5,2 | 0.0137 (0.00726) | 0.0078 (0.00349) | 0.0110 (0.00424)
  Days 8 to 10: n=6,6,2 | 0.0178 (0.01139) | 0.0088 (0.00264) | 0.0130 (0.00424)

50. Secondary Outcome: Part 2: Absolute Values for Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Leukocytes, Platelet Count
Description: Blood samples were collected to analyze the hematology parameters: basophils, eosinophils, lymphocytes, monocytes, neutrophils, leukocytes and platelet count. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
10^9 cells per liter
  Baseline (Day 1): Basophils, n=6,6,5,2: number analyzed (Participants) | 6 | 6 | 5 | 2
  Baseline (Day 1): Basophils, n=6,6,5,2 | 0.042 (0.0232) | 0.042 (0.0117) | 0.030 (0.0200) | 0.040 (0.0283)
  Day 7: Basophils, n=5,6,5,2: number analyzed (Participants) | 5 | 6 | 5 | 2
  Day 7: Basophils, n=5,6,5,2 | 0.050 (0.0274) | 0.062 (0.0223) | 0.054 (0.0251) | 0.035 (0.0071)
  Baseline (Day 1): Eosinophils, n=6,6,5,2: number analyzed (Participants) | 6 | 6 | 5 | 2
  Baseline (Day 1): Eosinophils, n=6,6,5,2 | 0.402 (0.3307) | 0.290 (0.2628) | 0.320 (0.2542) | 0.055 (0.0354)
  Day 7: Eosinophils, n=5,6,5,2: number analyzed (Participants) | 5 | 6 | 5 | 2
  Day 7: Eosinophils, n=5,6,5,2 | 0.316 (0.1780) | 0.243 (0.1546) | 0.210 (0.1239) | 0.075 (0.0354)
  Baseline (Day 1): Lymphocytes, n=6,6,5,2: number analyzed (Participants) | 6 | 6 | 5 | 2
  Baseline (Day 1): Lymphocytes, n=6,6,5,2 | 1.990 (0.3013) | 2.047 (0.6167) | 2.236 (0.3010) | 1.865 (0.3606)
  Day 7: Lymphocytes, n=5,6,5,2: number analyzed (Participants) | 5 | 6 | 5 | 2
  Day 7: Lymphocytes, n=5,6,5,2 | 1.960 (0.3450) | 1.985 (0.2983) | 2.694 (0.7060) | 1.755 (0.0919)
  Baseline (Day 1): Monocytes, n=6,6,5,2: number analyzed (Participants) | 6 | 6 | 5 | 2
  Baseline (Day 1): Monocytes, n=6,6,5,2 | 0.560 (0.2082) | 0.477 (0.1442) | 0.534 (0.1459) | 0.435 (0.1061)
  Day 7: Monocytes, n=5,6,5,2: number analyzed (Participants) | 5 | 6 | 5 | 2
  Day 7: Monocytes, n=5,6,5,2 | 0.530 (0.2210) | 0.498 (0.2647) | 0.414 (0.1467) | 0.305 (0.0071)
  Baseline (Day 1): Neutrophils, n=6,6,5,2: number analyzed (Participants) | 6 | 6 | 5 | 2
  Baseline (Day 1): Neutrophils, n=6,6,5,2 | 2.512 (1.2631) | 2.442 (1.1951) | 3.060 (0.5711) | 2.280 (1.0465)
  Day 7: Neutrophils, n=5,6,5,2: number analyzed (Participants) | 5 | 6 | 5 | 2
  Day 7: Neutrophils, n=5,6,5,2 | 2.826 (1.1821) | 4.120 (2.9025) | 3.344 (0.6322) | 2.065 (1.3647)
  Baseline (Day 1): Leukocytes, n=6,6,5,2: number analyzed (Participants) | 6 | 6 | 5 | 2
  Baseline (Day 1): Leukocytes, n=6,6,5,2 | 5.50 (1.633) | 5.28 (1.947) | 6.20 (0.938) | 4.65 (1.485)
  Day 7: Leukocytes, n=5,6,6,2: number analyzed (Participants) | 5 | 6 | 6 | 2
  Day 7: Leukocytes, n=5,6,6,2 | 5.66 (1.527) | 6.90 (3.310) | 6.55 (0.973) | 4.20 (1.414)
  Baseline (Day 1): Platelet count, n=5,6,5,2: number analyzed (Participants) | 5 | 6 | 5 | 2
  Baseline (Day 1): Platelet count, n=5,6,5,2 | 276.6 (54.29) | 236.7 (41.87) | 232.2 (40.12) | 197.0 (59.40)
  Day 7: Platelet count, n=4,6,6,2: number analyzed (Participants) | 4 | 6 | 6 | 2
  Day 7: Platelet count, n=4,6,6,2 | 292.0 (77.06) | 254.2 (37.39) | 249.0 (38.72) | 201.5 (60.10)

51. Secondary Outcome: Part 2: Absolute Values for Hematology Parameter: Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Grams per liter
  Baseline (Day 1): n=6,6,5,2: number analyzed (Participants) | 6 | 6 | 5 | 2
  Baseline (Day 1): n=6,6,5,2 | 136.3 (16.34) | 149.2 (13.44) | 141.2 (7.98) | 147.0 (7.07)
  Day 7: n=5,6,6,2: number analyzed (Participants) | 5 | 6 | 6 | 2
  Day 7: n=5,6,6,2 | 129.4 (19.55) | 144.5 (7.87) | 135.8 (11.02) | 139.0 (8.49)

52. Secondary Outcome: Part 2: Absolute Values for Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Proportion of red blood cells in blood
  Baseline (Day 1): n=6,6,5,2: number analyzed (Participants) | 6 | 6 | 5 | 2
  Baseline (Day 1): n=6,6,5,2 | 0.4037 (0.04646) | 0.4505 (0.02992) | 0.4222 (0.01879) | 0.4330 (0.01838)
  Day 7: n=5,6,6,2: number analyzed (Participants) | 5 | 6 | 6 | 2
  Day 7: n=5,6,6,2 | 0.3826 (0.05125) | 0.4382 (0.01579) | 0.4062 (0.03107) | 0.4015 (0.03323)

53. Secondary Outcome: Part 2: Absolute Values for Hematology Parameter: Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
10^12 cells per liter
  Baseline (Day 1): n=6,6,5,2: number analyzed (Participants) | 6 | 6 | 5 | 2
  Baseline (Day 1): n=6,6,5,2 | 4.53 (0.476) | 5.17 (0.450) | 4.74 (0.230) | 4.80 (0.000)
  Day 7: n=5,6,6,2: number analyzed (Participants) | 5 | 6 | 6 | 2
  Day 7: n=5,6,6,2 | 4.26 (0.503) | 5.00 (0.518) | 4.52 (0.431) | 4.50 (0.000)

54. Secondary Outcome: Part 2: Absolute Values for Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular volume. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Femtoliter
  Baseline (Day 1): n=6,6,5,2: number analyzed (Participants) | 6 | 6 | 5 | 2
  Baseline (Day 1): n=6,6,5,2 | 88.8 (3.76) | 87.8 (8.59) | 89.2 (1.64) | 91.0 (4.24)
  Day 7: n=5,6,6,2: number analyzed (Participants) | 5 | 6 | 6 | 2
  Day 7: n=5,6,6,2 | 89.6 (3.44) | 88.0 (8.53) | 90.0 (2.97) | 89.0 (7.07)

55. Secondary Outcome: Part 2: Absolute Values for Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Picograms
  Baseline (Day 1): n=6,6,5,2: number analyzed (Participants) | 6 | 6 | 5 | 2
  Baseline (Day 1): n=6,6,5,2 | 30.07 (1.870) | 29.15 (3.531) | 29.80 (0.925) | 30.95 (1.485)
  Day 7: n=5,6,6,2: number analyzed (Participants) | 5 | 6 | 6 | 2
  Day 7: n=5,6,6,2 | 30.22 (2.017) | 29.10 (3.553) | 29.97 (0.898) | 30.90 (1.838)

56. Secondary Outcome: Part 2: Absolute Values for Hematology Parameter: Reticulocytes/Erythro
Description: Blood samples were collected to analyze the hematology parameter: reticulocytes/erythro. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percentage of reticulocytes in erythro
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Percentage of reticulocytes in erythro
  Baseline (Day 1): n=6,6,5,2: number analyzed (Participants) | 6 | 6 | 5 | 2
  Baseline (Day 1): n=6,6,5,2 | 0.0102 (0.00223) | 0.0082 (0.00147) | 0.0108 (0.00492) | 0.0070 (0.00141)
  Day 7: n=5,6,6,2: number analyzed (Participants) | 5 | 6 | 6 | 2
  Day 7: n=5,6,6,2 | 0.0124 (0.00297) | 0.0098 (0.00160) | 0.0107 (0.00344) | 0.0090 (0.00141)

57. Secondary Outcome: Part 1: Absolute Values for Chemistry Parameters: Glucose, Cholesterol, Triglycerides, Calcium, Chloride, Phosphate, Potassium, Magnesium, Sodium, Urea, HDL Cholesterol, LDL Cholesterol
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the chemistry parameters: glucose, cholesterol, triglycerides, calcium, chloride, phosphate, potassium, magnesium, sodium, urea, HDL cholesterol and LDL cholesterol. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Millimoles per liter
  Baseline (Day 1): Glucose, n=6,6,2 | 5.28 (0.556) | 4.88 (0.546) | 5.40 (0.141)
  Days 8 to 10: Glucose, n=6,6,2 | 5.08 (0.618) | 5.17 (0.528) | 5.40 (0.283)
  Baseline (Day 1): Cholesterol, n=6,6,2 | 4.700 (1.2345) | 4.058 (0.9641) | 4.350 (0.6364)
  Days 8 to 10: Cholesterol, n=0,0,0: number analyzed (Participants) | 0 | 0 | 0
  Baseline (Day 1): Triglycerides, n=6,6,2 | 1.070 (0.4527) | 1.150 (0.5114) | 0.950 (0.4101)
  Days 8 to 10: Triglycerides, n=0,0,0: number analyzed (Participants) | 0 | 0 | 0
  Baseline (Day 1): Calcium, n=6,6,2 | 2.300 (0.1073) | 2.313 (0.0961) | 2.330 (0.0141)
  Days 8 to 10: Calcium, n=6,6,2 | 2.293 (0.0816) | 2.287 (0.0561) | 2.350 (0.0424)
  Baseline (Day 1): Chloride, n=6,6,2 | 104.2 (0.41) | 105.8 (2.48) | 105.0 (2.83)
  Days 8 to 10: Chloride, n=6,6,2 | 104.2 (1.72) | 106.7 (1.21) | 104.5 (0.71)
  Baseline (Day 1): Phosphate, n=6,6,2 | 1.117 (0.1835) | 1.083 (0.1889) | 1.200 (0.0707)
  Days 8 to 10: Phosphate, n=6,6,2 | 1.158 (0.1882) | 1.142 (0.2245) | 1.125 (0.1768)
  Baseline (Day 1): Potassium, n=6,6,2 | 4.10 (0.210) | 4.30 (0.276) | 4.15 (0.212)
  Days 8 to 10: Potassium, n=6,6,2 | 4.12 (0.349) | 4.27 (0.216) | 4.05 (0.212)
  Baseline (Day 1): Magnesium, n=6,6,2 | 0.847 (0.0393) | 0.853 (0.0450) | 0.880 (0.0283)
  Days 8 to 10: Magnesium, n=6,6,2 | 0.847 (0.0561) | 0.847 (0.0393) | 0.860 (0.0000)
  Baseline (Day 1): Sodium, n=6,6,2 | 138.3 (2.25) | 139.8 (0.75) | 139.0 (0.00)
  Days 8 to 10: Sodium, n=6,6,2 | 138.5 (2.17) | 139.0 (0.89) | 138.0 (1.41)
  Baseline (Day 1): Urea, n=6,6,2 | 5.33 (0.516) | 5.83 (1.169) | 5.00 (0.707)
  Days 8 to 10: Urea, n=6,6,2 | 5.25 (1.037) | 5.75 (0.524) | 6.00 (0.707)
  Baseline (Day 1): HDL cholesterol, n=6,6,2 | 1.192 (0.1960) | 1.025 (0.0612) | 1.075 (0.0354)
  Days 8 to 10: HDL cholesterol, n=0,0,0: number analyzed (Participants) | 0 | 0 | 0
  Baseline (Day 1): LDL cholesterol, n=6,6,2 | 3.017 (1.0452) | 2.507 (0.7842) | 2.840 (0.4808)
  Days 8 to 10: LDL cholesterol, n=0,0,0: number analyzed (Participants) | 0 | 0 | 0

58. Secondary Outcome: Part 1: Absolute Values for Chemistry Parameters: ALT, ALP, AST
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the chemistry parameters: ALT, ALP and AST. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
International units per liter
  Baseline (Day 1): ALT | 31.3 (15.67) | 19.7 (15.82) | 20.0 (8.49)
  Days 8 to 10: ALT | 34.0 (21.58) | 18.0 (11.85) | 29.5 (14.85)
  Baseline (Day 1): ALP | 62.0 (10.55) | 62.3 (19.13) | 63.0 (2.83)
  Days 8 to 10: ALP | 72.5 (27.68) | 58.8 (16.46) | 59.0 (1.41)
  Baseline (Day 1): AST | 26.7 (9.42) | 23.3 (10.76) | 20.0 (8.49)
  Days 8 to 10: AST | 26.2 (11.27) | 21.3 (4.63) | 24.5 (10.61)

59. Secondary Outcome: Part 1: Absolute Values for Chemistry Parameters: Creatinine, Bilirubin
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the chemistry parameters: creatinine and bilirubin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Micromoles per liter
  Baseline (Day 1): Creatinine | 82.05 (11.319) | 81.35 (3.861) | 88.40 (3.818)
  Days 8 to 10: Creatinine | 83.82 (13.674) | 80.02 (6.239) | 88.40 (3.818)
  Baseline (Day 1): Bilirubin | 11.7 (6.38) | 8.0 (2.83) | 15.0 (1.41)
  Days 8 to 10: Bilirubin | 11.3 (3.50) | 6.0 (1.79) | 18.0 (8.49)

60. Secondary Outcome: Part 1: Absolute Values for Chemistry Parameters: Protein
Description: Blood samples were collected at Baseline and one sample between Days 8 to 10 to analyze the chemistry parameter: protein. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Grams per liter
  Baseline (Day 1) | 72.2 (3.06) | 70.3 (2.34) | 69.0 (1.41)
  Days 8 to 10 | 70.8 (3.60) | 69.3 (5.05) | 70.0 (1.41)

61. Secondary Outcome: Part 1: Absolute Values for Chemistry Parameters: Amylase, Lipase
Description: Blood samples were collected to analyze the chemistry parameters: amylase and lipase. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 6 (Day 11)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 2 | 0 | 0
Units per liter
  Baseline (Day 1): Amylase | 57.0 (11.31) |  |
  Day 11: Amylase | 57.0 (0.00) |  |
  Baseline (Day 1): Lipase | 28.5 (4.95) |  |
  Day 11: Lipase | 26.5 (7.78) |  |

62. Secondary Outcome: Part 2: Absolute Values for Chemistry Parameters: Glucose, Cholesterol, Triglycerides, Calcium, Chloride, Phosphate, Potassium, Magnesium, Sodium, Urea, HDL Cholesterol, LDL Cholesterol
Description: Blood samples were collected to analyze the chemistry parameters: glucose, cholesterol, triglycerides, calcium, chloride, phosphate, potassium, magnesium, sodium, urea, HDL cholesterol and LDL cholesterol. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Millimoles per liter
  Baseline (Day 1): Glucose, n=6,6,6,2 | 4.68 (0.306) | 4.72 (0.928) | 4.80 (0.456) | 4.90 (0.849)
  Day 7: Glucose, n=6,6,6,1: number analyzed (Participants) | 6 | 6 | 6 | 1
  Day 7: Glucose, n=6,6,6,1 | 4.63 (0.408) | 4.90 (0.190) | 4.77 (0.320) | 4.80 (NA) — Standard deviation could not be calculated for single participant.
  Baseline (Day 1): Cholesterol, n=6,6,6,2 | 4.233 (0.6758) | 4.375 (1.1626) | 4.150 (0.8573) | 3.400 (0.3536)
  Day 7: Cholesterol, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Baseline (Day 1): Triglycerides, n=6,6,6,2 | 1.183 (0.1924) | 1.447 (0.6008) | 1.120 (0.4879) | 0.540 (0.1980)
  Day 7: Triglycerides, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Baseline (Day 1): Calcium, n=6,6,6,2 | 2.330 (0.0629) | 2.320 (0.0980) | 2.290 (0.0701) | 2.280 (0.0849)
  Day 7: Calcium, n=6,6,6,1: number analyzed (Participants) | 6 | 6 | 6 | 1
  Day 7: Calcium, n=6,6,6,1 | 2.273 (0.0628) | 2.293 (0.0766) | 2.320 (0.0780) | 2.220 (NA) — Standard deviation could not be calculated for single participant.
  Baseline (Day 1): Chloride, n=6,6,6,2 | 103.0 (1.67) | 102.2 (2.64) | 103.7 (2.34) | 105.5 (0.71)
  Day 7: Chloride, n=6,6,6,1: number analyzed (Participants) | 6 | 6 | 6 | 1
  Day 7: Chloride, n=6,6,6,1 | 102.3 (1.51) | 102.0 (1.79) | 103.0 (1.10) | 104.0 (NA) — Standard deviation could not be calculated for single participant.
  Baseline (Day 1): Phosphate, n=6,6,6,2 | 1.317 (0.1693) | 1.108 (0.1281) | 1.083 (0.1211) | 0.950 (0.2828)
  Day 7: Phosphate, n=6,6,6,1: number analyzed (Participants) | 6 | 6 | 6 | 1
  Day 7: Phosphate, n=6,6,6,1 | 1.200 (0.1265) | 1.175 (0.1969) | 1.167 (0.1329) | 0.750 (NA) — Standard deviation could not be calculated for single participant.
  Baseline (Day 1): Potassium, n=6,6,6,2 | 4.07 (0.476) | 3.98 (0.325) | 3.95 (0.164) | 4.10 (0.424)
  Day 7: Potassium, n=6,6,6,1: number analyzed (Participants) | 6 | 6 | 6 | 1
  Day 7: Potassium, n=6,6,6,1 | 3.87 (0.273) | 4.03 (0.242) | 4.15 (0.122) | 3.70 (NA) — Standard deviation could not be calculated for single participant.
  Baseline (Day 1): Magnesium, n=6,6,6,2 | 0.790 (0.0395) | 0.830 (0.0518) | 0.803 (0.0320) | 0.810 (0.0707)
  Day 7: Magnesium, n=6,6,6,1: number analyzed (Participants) | 6 | 6 | 6 | 1
  Day 7: Magnesium, n=6,6,6,1 | 0.797 (0.0731) | 0.837 (0.0427) | 0.830 (0.0654) | 0.760 (NA) — Standard deviation could not be calculated for single participant.
  Baseline (Day 1): Sodium, n=6,6,6,2 | 137.7 (1.63) | 138.5 (2.43) | 137.8 (3.06) | 140.5 (2.12)
  Day 7: Sodium, n=6,6,6,1: number analyzed (Participants) | 6 | 6 | 6 | 1
  Day 7: Sodium, n=6,6,6,1 | 136.8 (3.54) | 138.2 (1.94) | 137.7 (1.97) | 138.0 (NA) — Standard deviation could not be calculated for single participant.
  Baseline (Day 1): Urea, n=6,6,6,2 | 4.50 (1.517) | 4.25 (1.508) | 5.92 (1.068) | 6.25 (2.475)
  Day 7: Urea, n=6,6,6,1: number analyzed (Participants) | 6 | 6 | 6 | 1
  Day 7: Urea, n=6,6,6,1 | 4.08 (0.970) | 4.00 (0.632) | 5.58 (0.492) | 4.00 (NA) — Standard deviation could not be calculated for single participant.
  Baseline (Day 1): HDL cholesterol, n=6,6,6,2 | 1.242 (0.3277) | 1.133 (0.3312) | 1.200 (0.3194) | 1.250 (0.0707)
  Day 7: HDL cholesterol, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0
  Baseline (Day 1): LDL cholesterol, n=6,6,6,2 | 2.448 (0.6649) | 2.578 (0.8267) | 2.437 (0.6955) | 1.905 (0.3748)
  Day 7: LDL cholesterol, n=0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0

63. Secondary Outcome: Part 2: Absolute Values for Chemistry Parameters: ALT, ALP, AST
Description: Blood samples were collected to analyze the chemistry parameters: ALT, ALP and AST. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
International units per liter
  Baseline (Day 1): ALT, n=6,6,6,2 | 18.3 (14.07) | 17.8 (7.63) | 33.2 (23.07) | 34.5 (6.36)
  Day 7: ALT, n=6,6,6,1: number analyzed (Participants) | 6 | 6 | 6 | 1
  Day 7: ALT, n=6,6,6,1 | 14.5 (7.66) | 16.7 (5.24) | 27.0 (18.00) | 29.0 (NA) — Standard deviation could not be calculated for single participant.
  Baseline (Day 1): ALP, n=6,6,6,2 | 63.3 (15.08) | 63.7 (4.68) | 60.8 (9.00) | 43.0 (18.38)
  Day 7: ALP, n=6,6,6,1: number analyzed (Participants) | 6 | 6 | 6 | 1
  Day 7: ALP, n=6,6,6,1 | 60.2 (16.53) | 63.0 (5.25) | 59.0 (5.18) | 55.0 (NA) — Standard deviation could not be calculated for single participant.
  Baseline (Day 1): AST, n=6,6,6,2 | 26.8 (15.39) | 18.5 (6.60) | 26.7 (8.14) | 50.0 (39.60)
  Day 7: AST, n=6,6,6,1: number analyzed (Participants) | 6 | 6 | 6 | 1
  Day 7: AST, n=6,6,6,1 | 21.7 (6.74) | 18.8 (3.31) | 22.0 (3.74) | 26.0 (NA) — Standard deviation could not be calculated for single participant.

64. Secondary Outcome: Part 2: Absolute Values for Chemistry Parameters: Creatinine, Bilirubin
Description: Blood samples were collected to analyze the chemistry parameters: creatinine and bilirubin. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Micromoles per liter
  Baseline (Day 1): Creatinine, n=6,6,6,2 | 71.30 (12.207) | 73.67 (7.120) | 73.52 (12.761) | 86.65 (13.789)
  Day 7: Creatinine, n=6,6,6,1: number analyzed (Participants) | 6 | 6 | 6 | 1
  Day 7: Creatinine, n=6,6,6,1 | 72.65 (14.109) | 70.28 (8.269) | 73.35 (8.195) | 76.00 (NA) — Standard deviation could not be calculated for single participant.
  Baseline (Day 1): Bilirubin, n=6,6,6,2 | 10.0 (5.66) | 9.3 (1.03) | 7.7 (3.44) | 11.0 (7.07)
  Day 7: Bilirubin, n=6,6,6,1: number analyzed (Participants) | 6 | 6 | 6 | 1
  Day 7: Bilirubin, n=6,6,6,1 | 9.7 (4.97) | 10.7 (5.47) | 8.0 (2.83) | 6.0 (NA) — Standard deviation could not be calculated for single participant.

65. Secondary Outcome: Part 2: Absolute Values for Chemistry Parameters: Protein
Description: Blood samples were collected to analyze the chemistry parameter: protein. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Grams per liter
  Baseline (Day 1): n=6,6,6,2 | 78.8 (12.78) | 73.3 (5.50) | 76.7 (10.03) | 73.5 (0.71)
  Day 7: n=6,6,6,1: number analyzed (Participants) | 6 | 6 | 6 | 1
  Day 7: n=6,6,6,1 | 76.7 (12.01) | 72.5 (5.13) | 78.2 (8.93) | 72.0 (NA) — Standard deviation could not be calculated for single participant.

66. Secondary Outcome: Part 2: Absolute Values for Chemistry Parameters: Amylase, Lipase
Description: as for outcome 61
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Units per liter
  Baseline (Day 1): Amylase, n=6,6,6,2 | 47.2 (18.15) | 51.0 (21.65) | 55.2 (18.61) | 56.0 (25.46)
  Day 7: Amylase, n=6,6,6,1: number analyzed (Participants) | 6 | 6 | 6 | 1
  Day 7: Amylase, n=6,6,6,1 | 44.8 (17.81) | 51.8 (22.71) | 61.8 (25.86) | 64.0 (NA) — Standard deviation could not be calculated for single participant.
  Baseline (Day 1): Lipase, n=6,6,6,2 | 26.5 (14.08) | 29.7 (10.95) | 43.2 (32.32) | 26.0 (14.14)
  Day 7: Lipase, n=6,6,6,1: number analyzed (Participants) | 6 | 6 | 6 | 1
  Day 7: Lipase, n=6,6,6,1 | 25.5 (11.64) | 27.5 (13.40) | 47.7 (34.70) | 44.0 (NA) — Standard deviation could not be calculated for single participant.

67. Secondary Outcome: Part 1: Absolute Values for Urinalysis Parameter: Specific Gravity
Description: Urine samples were collected at Baseline and one sample between Days 8 to 10 to analyze the urinalysis parameter: specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Ratio
  Baseline (Day 1) | 1.0238 (0.00677) | 1.0233 (0.00320) | 1.0240 (0.00283)
  Days 8 to 10 | 1.0240 (0.00533) | 1.0242 (0.00279) | 1.0240 (0.00000)

68. Secondary Outcome: Part 1: Absolute Values for Urinalysis Parameter: Urobilinogen
Description: Urine samples were collected at Baseline and one sample between Days 8 to 10 to analyze the urinalysis parameter: urobilinogen. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Micromoles per liter
  Baseline (Day 1) | 3.40 (0.000) | 3.40 (0.000) | 3.40 (0.000)
  Days 8 to 10 | 7.90 (6.971) | 3.40 (0.000) | 3.40 (0.000)

69. Secondary Outcome: Part 1: Absolute Values for Urinalysis Parameter: pH
Description: Urine samples were collected at Baseline and one sample between Days 8 to 10 to analyze the urinalysis parameter: pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acidic pH (5.0 - 6.0). Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
pH
  Baseline (Day 1) | 5.67 (0.931) | 5.75 (0.689) | 5.75 (0.354)
  Days 8 to 10 | 5.83 (0.753) | 5.42 (0.585) | 5.25 (0.354)

70. Secondary Outcome: Part 2: Absolute Values for Urinalysis Parameter: Specific Gravity
Description: Urine samples were collected to analyze the urinalysis parameter: specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Ratio
  Baseline (Day 1) | 1.0223 (0.00866) | 1.0272 (0.00360) | 1.0255 (0.00918) | 1.0375 (0.00495)
  Day 7 | 1.0233 (0.00686) | 1.0250 (0.00522) | 1.0273 (0.00327) | 1.0265 (0.00919)

71. Secondary Outcome: Part 2: Absolute Values for Urinalysis Parameter: Urobilinogen
Description: Urine samples were collected to analyze the urinalysis parameter: urobilinogen. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Micromoles per liter
  Baseline (Day 1) | 3.40 (0.000) | 3.40 (0.000) | 3.40 (0.000) | 3.40 (0.000)
  Day 7 | 3.40 (0.000) | 7.90 (6.971) | 3.40 (0.000) | 3.40 (0.000)

72. Secondary Outcome: Part 2: Absolute Values for Urinalysis Parameter: pH
Description: Urine samples were collected to analyze the urinalysis parameter: pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acidic pH (5.0 - 6.0). Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
pH
  Baseline (Day 1) | 5.33 (0.258) | 5.83 (0.753) | 5.25 (0.418) | 5.50 (0.000)
  Day 7 | 5.50 (0.775) | 5.67 (0.258) | 5.33 (0.258) | 5.75 (0.354)

73. Secondary Outcome: Part 1: Absolute Values for SBP and DBP
Description: SBP and DBP were measured in the semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Millimeters of mercury
  Baseline (Day 1): SBP | 120.2 (13.36) | 121.8 (12.25) | 106.0 (11.31)
  Days 8 to 10: SBP | 117.7 (8.87) | 122.3 (7.94) | 104.5 (7.78)
  Baseline (Day 1): DBP | 70.3 (17.32) | 66.7 (10.80) | 64.0 (5.66)
  Days 8 to 10: DBP | 70.0 (6.81) | 67.5 (9.91) | 64.5 (4.95)

74. Secondary Outcome: Part 1: Absolute Values for Respiratory Rate
Description: Respiratory rate was measured in the semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Breaths per minute
  Baseline (Day 1) | 16.0 (2.61) | 16.2 (3.31) | 15.0 (4.24)
  Days 8 to 10 | 15.0 (1.26) | 16.3 (2.73) | 14.0 (2.83)

75. Secondary Outcome: Part 1: Absolute Values for Pulse Rate
Description: Pulse rate was measured in the semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and Visit 5 (Days 8 to 10)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Beats per minute
  Baseline (Day 1) | 81.8 (18.25) | 65.8 (14.22) | 60.0 (2.83)
  Days 8 to 10 | 76.7 (21.13) | 71.3 (11.93) | 66.0 (5.66)

76. Secondary Outcome: Part 2: Absolute Values for SBP and DBP
Description: as for outcome 73
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Millimeters of mercury
  Baseline (Day 1): SBP | 117.0 (7.95) | 116.5 (11.04) | 112.2 (9.93) | 105.5 (2.12)
  Day 7: SBP | 118.0 (12.07) | 114.3 (8.36) | 119.5 (8.87) | 106.5 (4.95)
  Baseline (Day 1): DBP | 71.5 (4.51) | 74.0 (4.69) | 71.8 (12.89) | 71.0 (12.73)
  Day 7: DBP | 69.7 (4.50) | 73.0 (5.06) | 74.2 (5.27) | 70.5 (4.95)

77. Secondary Outcome: Part 2: Absolute Values for Respiratory Rate
Description: as for outcome 74
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Breaths per minute
  Baseline (Day 1) | 17.3 (2.66) | 17.2 (1.17) | 17.2 (2.40) | 16.0 (0.00)
  Day 7 | 17.2 (2.56) | 17.3 (2.07) | 16.2 (2.23) | 16.5 (2.12)

78. Secondary Outcome: Part 2: Absolute Values for Pulse Rate
Description: as for outcome 75
Time Frame: Baseline (Day 1) and Visit 5 (Day 7)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Beats per minute
  Baseline (Day 1) | 68.3 (9.91) | 74.5 (8.36) | 77.0 (10.16) | 64.5 (13.44)
  Day 7 | 72.5 (16.34) | 76.5 (7.87) | 79.8 (12.45) | 75.0 (5.66)

79. Secondary Outcome: Part 1: Absolute Values for ECG Parameters: PR, QRS, QT, QTcB and QTcF Intervals
Description: Twelve lead ECGs were obtained to measure PR interval, QRS duration, QT interval, QTcF interval and QTcB interval. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1), Visit 5 (Days 8 to 10: Pre-dose, 2, 4 and 6 hours)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo
Number analyzed (Participants) | 6 | 6 | 2
Milliseconds
  PR Interval- Baseline (Day 1) | 136.6 (14.49) | 168.4 (15.48) | 176.5 (27.58)
  PR Interval- Days 8 to 10: Pre-dose | 136.2 (15.26) | 160.8 (19.60) | 174.0 (29.70)
  PR Interval- Days 8 to 10: 2 hours | 138.0 (14.46) | 162.2 (11.53) | 165.0 (28.28)
  PR Interval- Days 8 to 10: 4 hours | 136.5 (12.10) | 168.7 (13.81) | 173.0 (28.28)
  PR Interval- Days 8 to 10: 6 hours | 138.0 (9.10) | 162.5 (15.06) | 151.5 (23.33)
  QRS Duration- Baseline (Day 1) | 93.1 (4.54) | 95.7 (6.85) | 85.8 (11.08)
  QRS Duration- Days 8 to 10: Pre-dose | 90.0 (7.46) | 92.3 (7.74) | 80.5 (7.78)
  QRS Duration- Days 8 to 10: 2 hours | 91.0 (6.36) | 96.2 (7.17) | 86.0 (7.07)
  QRS Duration- Days 8 to 10: 4 hours | 89.8 (5.91) | 94.0 (6.42) | 84.5 (14.85)
  QRS Duration- Days 8 to 10: 6 hours | 89.5 (7.04) | 92.8 (10.11) | 83.5 (2.12)
  QT Interval- Baseline (Day 1) | 367.6 (26.04) | 378.7 (26.75) | 372.7 (29.70)
  QT Interval- Days 8 to 10: Pre-dose | 368.3 (23.35) | 376.0 (31.46) | 353.0 (8.49)
  QT Interval- Days 8 to 10: 2 hours | 365.2 (25.39) | 383.2 (26.84) | 344.0 (25.46)
  QT Interval- Days 8 to 10: 4 hours | 376.3 (22.70) | 387.7 (29.34) | 347.5 (10.61)
  QT Interval- Days 8 to 10: 6 hours | 373.3 (26.48) | 384.5 (25.37) | 348.5 (7.78)
  QTcB Interval- Baseline (Day 1) | 412.15 (31.539) | 397.75 (22.914) | 388.43 (39.598)
  QTcB Interval- Days 8 to 10: Pre-dose | 413.80 (42.176) | 401.35 (22.923) | 387.05 (33.163)
  QTcB Interval- Days 8 to 10: 2 hours | 401.70 (37.316) | 393.15 (26.290) | 361.05 (7.283)
  QTcB Interval- Days 8 to 10: 4 hours | 412.92 (42.143) | 387.38 (24.454) | 358.20 (12.162)
  QTcB Interval- Days 8 to 10: 6 hours | 414.80 (34.569) | 388.60 (23.893) | 383.55 (28.496)
  QTcF Interval- Baseline (Day 1) | 396.2 (17.67) | 391.2 (19.11) | 383.2 (36.06)
  QTcF Interval- Days 8 to 10: Pre-dose | 397.3 (25.34) | 392.3 (20.64) | 375.5 (24.75)
  QTcF Interval- Days 8 to 10: 2 hours | 388.7 (22.72) | 389.8 (22.89) | 355.5 (13.44)
  QTcF Interval- Days 8 to 10: 4 hours | 399.8 (25.87) | 387.5 (21.27) | 354.5 (4.95)
  QTcF Interval- Days 8 to 10: 6 hours | 400.2 (19.22) | 387.3 (22.03) | 371.0 (21.21)

80. Secondary Outcome: Part 2: Absolute Values for ECG Parameters: PR, QRS, QT, QTcB and QTcF Intervals
Description: as for outcome 79
Time Frame: Baseline (Day 1), Visit 5 (Day 7: Pre-dose, 2, 4 and 6 hours)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 2
Milliseconds
  PR Interval- Baseline (Day 1) | 156.8 (33.02) | 162.9 (29.73) | 162.8 (20.83) | 144.3 (6.13)
  PR Interval- Day 7: Pre-dose | 166.5 (25.62) | 161.8 (31.06) | 155.5 (26.10) | 137.0 (5.66)
  PR Interval- Day 7: 2 hours | 162.8 (28.34) | 160.5 (28.73) | 159.7 (26.04) | 150.5 (3.54)
  PR Interval- Day 7: 4 hours | 162.0 (24.85) | 164.0 (31.51) | 154.5 (20.51) | 149.0 (11.31)
  PR Interval- Day 7: 6 hours | 160.7 (24.81) | 160.7 (27.25) | 160.7 (25.90) | 136.5 (3.54)
  QRS Duration- Baseline (Day 1) | 92.6 (10.22) | 95.1 (21.97) | 88.9 (7.40) | 85.7 (11.31)
  QRS Duration- Day 7: Pre-dose | 96.5 (8.14) | 98.3 (28.86) | 88.5 (3.99) | 88.0 (4.24)
  QRS Duration- Day 7: 2 hours | 95.0 (9.78) | 95.8 (19.29) | 88.8 (4.49) | 90.0 (12.73)
  QRS Duration- Day 7: 4 hours | 94.3 (8.89) | 95.2 (18.94) | 85.8 (4.88) | 89.5 (7.78)
  QRS Duration- Day 7: 6 hours | 93.2 (10.61) | 95.0 (21.29) | 88.2 (8.11) | 88.5 (17.68)
  QT Interval- Baseline (Day 1) | 386.6 (28.86) | 355.9 (25.37) | 362.5 (19.45) | 378.8 (1.18)
  QT Interval- Day 7: Pre-dose | 379.2 (33.30) | 354.3 (31.94) | 367.5 (26.93) | 382.0 (1.41)
  QT Interval- Day 7: 2 hours | 362.2 (31.24) | 351.5 (25.05) | 364.3 (17.32) | 378.5 (4.95)
  QT Interval- Day 7: 4 hours | 373.8 (24.25) | 360.2 (23.07) | 360.8 (18.64) | 390.0 (18.38)
  QT Interval- Day 7: 6 hours | 365.2 (34.53) | 361.8 (25.88) | 363.2 (19.50) | 381.5 (6.36)
  QTcB Interval- Baseline (Day 1) | 402.88 (26.814) | 398.24 (25.587) | 411.18 (15.858) | 406.73 (20.742)
  QTcB Interval- Day 7: Pre-dose | 398.72 (26.663) | 398.58 (21.075) | 414.63 (17.816) | 399.65 (18.173)
  QTcB Interval- Day 7: 2 hours | 405.78 (10.923) | 398.33 (33.672) | 406.30 (27.565) | 388.50 (17.819)
  QTcB Interval- Day 7: 4 hours | 395.92 (22.851) | 397.68 (20.635) | 412.48 (27.377) | 382.90 (17.961)
  QTcB Interval- Day 7: 6 hours | 399.62 (19.074) | 402.42 (22.916) | 409.50 (19.009) | 396.90 (3.253)
  QTcF Interval- Baseline (Day 1) | 397.4 (24.60) | 383.5 (23.72) | 394.1 (12.71) | 397.3 (13.67)
  QTcF Interval- Day 7: Pre-dose | 391.5 (24.01) | 383.0 (24.90) | 398.2 (18.58) | 394.0 (12.73)
  QTcF Interval- Day 7: 2 hours | 390.2 (12.16) | 382.2 (30.20) | 391.8 (22.44) | 385.0 (14.14)
  QTcF Interval- Day 7: 4 hours | 388.0 (18.21) | 384.7 (20.42) | 394.7 (18.91) | 385.0 (18.38)
  QTcF Interval- Day 7: 6 hours | 387.8 (11.29) | 388.0 (21.76) | 393.3 (17.20) | 391.5 (4.95)

81. Secondary Outcome: Part 1: Area Under the Plasma Concentration Time Curve From Zero to 24 (AUC[0-24]) Following Administration of GSK3640254 on Day 1
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3640254. The PK parameters were calculated by standard non-compartmental analysis. Pharmacokinetic (PK) Population consisted of all participants who received GSK3640254 and underwent plasma PK sampling during the study.
Time Frame: Day 1: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg
Number analyzed (Participants) | 5 | 6
Hours*microgram per milliliter | 0.6946 (13.5) | 12.3929 (91.3)

82. Secondary Outcome: Part 1: Maximum Observed Concentration (Cmax) Following Administration of GSK3640254 on Day 1
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3640254. The PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Day 1: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg
Number analyzed (Participants) | 6 | 6
Microgram per milliliter | 0.0591 (177.4) | 0.9381 (82.3)

83. Secondary Outcome: Part 1: Time to Maximum Observed Concentration (Tmax) Following Administration of GSK3640254 on Day 1
Description: as for outcome 82
Time Frame: Day 1: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg
Number analyzed (Participants) | 6 | 6
Hours | 2.9250 [0.000 to 5.000] | 5.5250 [3.917 to 8.050]

84. Secondary Outcome: Part 1: Concentration at 24 Hours Post-dose (C24) Following Administration of GSK3640254 on Day 1
Description: as for outcome 82
Time Frame: Day 1: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg
Number analyzed (Participants) | 6 | 6
Microgram per milliliter | 0.0180 (27.5) | 0.3553 (92.7)

85. Secondary Outcome: Part 1: Absorption Lag Time (Tlag) Following Administration of GSK3640254 on Day 1
Description: as for outcome 82
Time Frame: Day 1: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg
Number analyzed (Participants) | 6 | 6
Hours | 0.500 [0.00 to 1.00] | 0.000 [0.00 to 1.00]

86. Secondary Outcome: Part 2: AUC(0-24) Following Administration of GSK3640254 on Day 1
Description: as for outcome 82
Time Frame: Day 1: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg
Number analyzed (Participants) | 6 | 6 | 6
Hours*microgram per milliliter | 3.2527 (31.7) | 6.1228 (38.8) | 14.0335 (36.6)

87. Secondary Outcome: Part 2: Cmax Following Administration of GSK3640254 on Day 1
Description: as for outcome 82
Time Frame: Day 1: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg
Number analyzed (Participants) | 6 | 6 | 6
Microgram per milliliter | 0.2316 (30.5) | 0.4329 (33.6) | 0.9178 (41.5)

88. Secondary Outcome: Part 2: Tmax Following Administration of GSK3640254 on Day 1
Description: as for outcome 82
Time Frame: Day 1: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg
Number analyzed (Participants) | 6 | 6 | 6
Hours | 4.4167 [3.967 to 8.000] | 4.0750 [2.950 to 6.167] | 5.5083 [3.000 to 6.250]

89. Secondary Outcome: Part 2: C24 Following Administration of GSK3640254 on Day 1
Description: as for outcome 82
Time Frame: Day 1: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg
Number analyzed (Participants) | 6 | 6 | 6
Microgram per milliliter | 0.0951 (33.7) | 0.1856 (36.2) | 0.4207 (33.8)

90. Secondary Outcome: Part 2: Tlag Following Administration of GSK3640254 on Day 1
Description: as for outcome 82
Time Frame: Day 1: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg
Number analyzed (Participants) | 6 | 6 | 6
Hours | 0.483 [0.00 to 2.00] | 0.000 [0.00 to 1.00] | 0.000 [0.00 to 1.00]

91. Secondary Outcome: Part 1: Area Under the Plasma Drug Concentration-time Curve From Pre-dose to the End of the Dosing Interval at Steady State (AUC[0-tau]) Following Repeat Dose Administration of GSK3640254 on Days 8 to 10
Description: as for outcome 82
Time Frame: Days 8 to 10: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg
Number analyzed (Participants) | 6 | 6
Hours*microgram per milliliter | 0.9082 (44.7) | 27.9363 (18.4)

92. Secondary Outcome: Part 1: Cmax Following Repeat Dose Administration of GSK3640254 on Days 8 to 10
Description: as for outcome 82
Time Frame: Days 8 to 10: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg
Number analyzed (Participants) | 6 | 6
Microgram per milliliter | 0.0549 (41.3) | 1.8559 (19.5)

93. Secondary Outcome: Part 1: Tmax Following Repeat Dose Administration of GSK3640254 on Days 8 to 10
Description: as for outcome 82
Time Frame: Days 8 to 10: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg
Number analyzed (Participants) | 6 | 6
Hours | 4.0167 [1.867 to 5.000] | 5.4833 [3.000 to 6.200]

94. Secondary Outcome: Part 1: Pre-dose Concentration (C0) Following Repeat Dose Administration of GSK3640254 on Days 8 to 10
Description: Blood sample was collected at indicated time point for pharmacokinetic analysis of GSK3640254. The PK parameters were calculated by standard non-compartmental analysis.
Time Frame: Days 8 to 10: Pre-dose
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg
Number analyzed (Participants) | 6 | 5
Microgram per milliliter | 0.0268 (41.6) | 0.6928 (33.6)

95. Secondary Outcome: Part 1: Concentration at End of Dosing Interval (Ctau) Following Repeat Dose Administration of GSK3640254 on Days 8 to 10
Description: as for outcome 82
Time Frame: Days 8 to 10: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg
Number analyzed (Participants) | 6 | 6
Microgram per milliliter | 0.0267 (47.0) | 0.7033 (29.6)

96. Secondary Outcome: Part 1: Apparent Terminal Phase Half-life (t1/2) Following Repeat Dose Administration of GSK3640254 on Days 8 to 10
Description: as for outcome 82
Time Frame: Days 8 to 10: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg
Number analyzed (Participants) | 6 | 6
Hours | NA [NA to NA] — t1/2 could not be calculated as the criteria of a span ratio [ratio of half-life to time used for half-life calculation] for at least 2 participants could not be fulfilled due to lack of available data. | NA [NA to NA] — t1/2 could not be calculated as the criteria of a span ratio [ratio of half-life to time used for half-life calculation] for at least 2 participants could not be fulfilled due to lack of available data.

97. Secondary Outcome: Part 1: Apparent Oral Clearance (CL/F) Following Repeat Dose Administration of GSK3640254 on Days 8 to 10
Description: as for outcome 82
Time Frame: Days 8 to 10: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter per hour
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg
Number analyzed (Participants) | 6 | 6
Milliliter per hour | 11010.5393 (44.7) | 7159.1443 (18.4)

98. Secondary Outcome: Part 2: AUC(0-tau) Following Repeat Dose Administration of GSK3640254 on Day 7
Description: as for outcome 82
Time Frame: Day 7: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg
Number analyzed (Participants) | 6 | 6 | 6
Hours*microgram per milliliter | 7.4626 (26.8) | 11.8256 (26.7) | 29.2952 (27.9)

99. Secondary Outcome: Part 2: Cmax Following Repeat Dose Administration of GSK3640254 on Day 7
Description: as for outcome 82
Time Frame: Day 7: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg
Number analyzed (Participants) | 6 | 6 | 6
Microgram per milliliter | 0.4692 (20.6) | 0.7470 (23.7) | 1.8574 (26.0)

100. Secondary Outcome: Part 2: Tmax Following Repeat Dose Administration of GSK3640254 on Day 7
Description: as for outcome 82
Time Frame: Day 7: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg
Number analyzed (Participants) | 6 | 6 | 6
Hours | 4.0583 [2.000 to 8.000] | 4.5750 [4.000 to 5.183] | 4.0750 [2.917 to 5.200]

101. Secondary Outcome: Part 2: C0 Following Repeat Dose Administration of GSK3640254 on Day 7
Description: as for outcome 94
Time Frame: Day 7: Pre-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg
Number analyzed (Participants) | 6 | 6 | 6
Microgram per milliliter | 0.2155 (24.2) | 0.3575 (38.0) | 0.7520 (38.8)

102. Secondary Outcome: Part 2: Ctau Following Repeat Dose Administration of GSK3640254 on Day 7
Description: as for outcome 82
Time Frame: Day 7: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg
Number analyzed (Participants) | 6 | 6 | 6
Microgram per milliliter | 0.2187 (30.1) | 0.3599 (31.1) | 0.7979 (34.1)

103. Secondary Outcome: Part 2: t1/2 Following Repeat Dose Administration of GSK3640254 on Day 7
Description: as for outcome 82
Time Frame: Day 7: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg
Number analyzed (Participants) | 6 | 6 | 6
Hours | NA [NA to NA] — t1/2 could not be calculated as the criteria of a span ratio [ratio of half-life to time used for half-life calculation] for at least 2 participants could not be fulfilled due to lack of available data. | NA [NA to NA] — t1/2 could not be calculated as the criteria of a span ratio [ratio of half-life to time used for half-life calculation] for at least 2 participants could not be fulfilled due to lack of available data. | NA [NA to NA] — t1/2 could not be calculated as the criteria of a span ratio [ratio of half-life to time used for half-life calculation] for at least 2 participants could not be fulfilled due to lack of available data.

104. Secondary Outcome: Part 2: CL/F Following Repeat Dose Administration of GSK3640254 on Day 7
Description: as for outcome 82
Time Frame: Day 7: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter per hour
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg
Number analyzed (Participants) | 6 | 6 | 6
Milliliter per hour | 5360.0526 (26.8) | 6764.9862 (26.7) | 4778.9430 (27.9)

105. Secondary Outcome: Part 1 and Part 2: Change From Baseline in Plasma HIV-1 RNA Relative to Day 8 AUC(0-tau)
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value. Statistical analysis for relationship between PK parameters (AUC) and PD measures (Change from Baseline in plasma HIV-1 RNA) were explored using a frequentist three parameter Emax non-linear model. The model parameters estimated included: maximum response (Emax), PK parameter value that attains 50 percent (%) of the maximal effect (EC50) and residual variability (s2e). PK/PD Population consisted of participants who met criteria for Per-Protocol and Pharmacokinetic Population analysis sets and who underwent PD sampling during the study.
Time Frame: Baseline (Day 1) and Day 8
Population: PK/PD Population.
Measure: Mean (Standard Deviation); unit: Copies per milliliter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Copies per milliliter | 12071.4 (42117.29) | -113331.4 (89475.00) | -48655.0 (26269.41) | -37904.3 (38814.54) | -64861.5 (83728.15)
Statistical Analysis 1: Comparison: Part 1: GSK3640254 10 mg vs Part 1: GSK3640254 200 mg vs Part 2: GSK3640254 40 mg vs Part 2: GSK3640254 80 mg vs Part 2: GSK3640254 140 mg; Test type: Other; Emax = -1.937, 95% CI 2-sided [-2.484 to -1.389]
Statistical Analysis 2: Comparison: Part 1: GSK3640254 10 mg vs Part 1: GSK3640254 200 mg vs Part 2: GSK3640254 40 mg vs Part 2: GSK3640254 80 mg vs Part 2: GSK3640254 140 mg; Test type: Other; EC50 = 7.094, 95% CI 2-sided [0.585 to 13.602]
Statistical Analysis 3: Comparison: Part 1: GSK3640254 10 mg vs Part 1: GSK3640254 200 mg vs Part 2: GSK3640254 40 mg vs Part 2: GSK3640254 80 mg vs Part 2: GSK3640254 140 mg; Test type: Other; s2e = 0.137, 95% CI 2-sided [0.062 to 0.212]

106. Secondary Outcome: Part 1 and Part 2: Change From Baseline in Plasma HIV-1 RNA Relative to Day 8 Cmax
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value. Statistical analysis for relationship between PK parameters (Cmax) and PD measures (Change from Baseline in plasma HIV-1 RNA) were explored using a frequentist three parameter Emax non-linear model. The model parameters estimated included: Emax, EC50 and s2e.
Time Frame: Baseline (Day 1) and Day 8
Population: PK/PD Population.
Measure: Mean (Standard Deviation); unit: Copies per milliliter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Copies per milliliter | 12071.4 (42117.29) | -113331.4 (89475.00) | -48655.0 (26269.41) | -37904.3 (38814.54) | -64861.5 (83728.15)
Statistical Analysis 1: Comparison: Part 1: GSK3640254 10 mg vs Part 1: GSK3640254 200 mg vs Part 2: GSK3640254 40 mg vs Part 2: GSK3640254 80 mg vs Part 2: GSK3640254 140 mg; Test type: Other; Emax = -1.929, 95% CI 2-sided [-2.479 to -1.379]
Statistical Analysis 2: Comparison: Part 1: GSK3640254 10 mg vs Part 1: GSK3640254 200 mg vs Part 2: GSK3640254 40 mg vs Part 2: GSK3640254 80 mg vs Part 2: GSK3640254 140 mg; Test type: Other; EC50 = 0.446, 95% CI 2-sided [0.030 to 0.861]
Statistical Analysis 3: Comparison: Part 1: GSK3640254 10 mg vs Part 1: GSK3640254 200 mg vs Part 2: GSK3640254 40 mg vs Part 2: GSK3640254 80 mg vs Part 2: GSK3640254 140 mg; Test type: Other; s2e = 0.139, 95% CI 2-sided [0.063 to 0.216]

107. Secondary Outcome: Part 1 and Part 2: Change From Baseline in Plasma HIV-1 RNA Relative to Day 8 Ctau
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the Baseline value from the post-dose visit value. Statistical analysis for relationship between PK parameters (Ctau) and PD measures (Change from Baseline in plasma HIV-1 RNA) were explored using a frequentist three parameter Emax non-linear model. The model parameters estimated included: Emax, EC50 and s2e.
Time Frame: Baseline (Day 1) and Day 8
Population: PK/PD Population.
Measure: Mean (Standard Deviation); unit: Copies per milliliter
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Copies per milliliter | 12071.4 (42117.29) | -113331.4 (89475.00) | -48655.0 (26269.41) | -37904.3 (38814.54) | -64861.5 (83728.15)
Statistical Analysis 1: Comparison: Part 1: GSK3640254 10 mg vs Part 1: GSK3640254 200 mg vs Part 2: GSK3640254 40 mg vs Part 2: GSK3640254 80 mg vs Part 2: GSK3640254 140 mg; Test type: Other; Emax = -1.926, 95% CI 2-sided [-2.498 to -1.354]
Statistical Analysis 2: Comparison: Part 1: GSK3640254 10 mg vs Part 1: GSK3640254 200 mg vs Part 2: GSK3640254 40 mg vs Part 2: GSK3640254 80 mg vs Part 2: GSK3640254 140 mg; Test type: Other; EC50 = 0.197, 95% CI 2-sided [0.007 to 0.386]
Statistical Analysis 3: Comparison: Part 1: GSK3640254 10 mg vs Part 1: GSK3640254 200 mg vs Part 2: GSK3640254 40 mg vs Part 2: GSK3640254 80 mg vs Part 2: GSK3640254 140 mg; Test type: Other; s2e = 0.144, 95% CI 2-sided [0.065 to 0.222]

108. Secondary Outcome: Part 1: Accumulation Ratio Following Repeat Dose Administration of GSK3640254
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3640254. The accumulation ratios (Ro) were calculated as Ro_AUC equal to (=) AUC(0-tau) Days 8 to 10 divided by (/) AUC(0-24) Day 1; Ro_Cmax=Cmax Days 8 to 10/Cmax Day 1; and Ro_Ctau=Ctau Days 8 to 10/C24 Day 1.
Time Frame: Day 1: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose; Days 8 to 10: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg
Number analyzed (Participants) | 6 | 6
Ratio
  Ro_AUC(0-tau), n=5,6: number analyzed (Participants) | 5 | 6
  Ro_AUC(0-tau), n=5,6 | 1.5352 (24.5) | 2.2542 (72.1)
  Ro_Cmax, n=6,6 | 0.9287 (171.7) | 1.9785 (69.4)
  Ro_Ctau, n=6,6 | 1.4790 (22.2) | 1.9796 (61.2)

109. Secondary Outcome: Part 2: Accumulation Ratio Following Repeat Dose Administration of GSK3640254
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3640254. The accumulation ratios (Ro) were calculated as Ro_AUC=AUC(0-tau) Day 7/AUC(0-24) Day 1; Ro_Cmax=Cmax Day 7/Cmax Day 1; and Ro_Ctau=Ctau Day 7/C24 Day 1.
Time Frame: Days 1 and 7: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg
Number analyzed (Participants) | 6 | 6 | 6
Ratio
  Ro_AUC(0-tau) | 2.2943 (11.2) | 1.9314 (18.6) | 2.0875 (29.2)
  Ro_Cmax | 2.0258 (24.4) | 1.7258 (17.6) | 2.0236 (37.5)
  Ro_Ctau | 2.2985 (6.4) | 1.9389 (20.8) | 1.8967 (16.0)

110. Secondary Outcome: Part 1 and Part 2: Dose Proportionality of GSK3640254 Administered on Day 1 Based on AUC(0-24)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3640254. The PK parameters were calculated by standard non-compartmental analysis. Dose proportionality was assessed using Power model with logarithm of dose as fixed effect. Slope and 90% confidence interval for the slope are presented.
Time Frame: Day 1: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Groups:
- GSK3640254 10 mg to 200 mg: In Part 1, participants received GSK3640254 10 mg, 200 mg, capsules, orally for 10 days and in Part 2, participants received GSK3640254 40 mg, 80 mg, 140 mg, capsules, orally for 7 days.
Arm/Group | GSK3640254 10 mg to 200 mg
Number analyzed (Participants) | 30
Slope of log dose | 1.018 [0.876 to 1.160]

111. Secondary Outcome: Part 1 and Part 2: Dose Proportionality of GSK3640254 Administered on Day 1 Based on Cmax
Description: as for outcome 110
Time Frame: Day 1: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Arm/Group | GSK3640254 10 mg to 200 mg
Number analyzed (Participants) | 30
Slope of log dose | 0.964 [0.774 to 1.154]

112. Secondary Outcome: Part 1 and Part 2: Dose Proportionality of GSK3640254 Administered on Day 1 Based on C24
Description: as for outcome 110
Time Frame: Day 1: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Arm/Group | GSK3640254 10 mg to 200 mg
Number analyzed (Participants) | 30
Slope of log dose | 1.061 [0.924 to 1.199]

113. Secondary Outcome: Part 1 and Part 2: Dose Proportionality of GSK3640254 Following Repeat Dose Administration Based on AUC(0-tau)
Description: as for outcome 110
Time Frame: Days 8 to 10: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose; Day 7: Pre-dose and 1, 2, 3, 4, 5, 6, 8, 12 and 24 hours post-dose
Population: PK Population.
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Arm/Group | GSK3640254 10 mg to 200 mg
Number analyzed (Participants) | 30
Slope of log dose | 1.179 [1.074 to 1.283]

114. Secondary Outcome: Part 1 and Part 2: Dose Proportionality of GSK3640254 Following Repeat Dose Administration Based on Cmax
Description: as for outcome 110
Time Frame: as for outcome 113
Population: PK Population.
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Arm/Group | GSK3640254 10 mg to 200 mg
Number analyzed (Participants) | 30
Slope of log dose | 1.204 [1.107 to 1.302]

115. Secondary Outcome: Part 1 and Part 2: Dose Proportionality of GSK3640254 Following Repeat Dose Administration Based on Ctau
Description: as for outcome 110
Time Frame: as for outcome 113
Population: PK Population.
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Arm/Group | GSK3640254 10 mg to 200 mg
Number analyzed (Participants) | 30
Slope of log dose | 1.137 [1.018 to 1.257]

ADVERSE EVENTS:
Time Frame: Part 1: up to Day 24; Part 2: up to Day 12
Description: Safety Population consisted of all participants who were enrolled into the study with documented evidence of having received at least 1 dose of randomized treatment.
Arm/Group | Part 1: GSK3640254 10 mg | Part 1: GSK3640254 200 mg | Part 1: Placebo | Part 2: GSK3640254 40 mg | Part 2: GSK3640254 80 mg | Part 2: GSK3640254 140 mg | Part 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/2 | 0/6 | 0/6 | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/2 | 0/6 | 0/6 | 1/6 | 0/2
Other Adverse Events (participants affected / at risk) | 3/6 | 5/6 | 0/2 | 5/6 | 4/6 | 4/6 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: GSK3640254 10 mg (N=6) | Part 1: GSK3640254 200 mg (N=6) | Part 1: Placebo (N=2) | Part 2: GSK3640254 40 mg (N=6) | Part 2: GSK3640254 80 mg (N=6) | Part 2: GSK3640254 140 mg (N=6) | Part 2: Placebo (N=2)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: GSK3640254 10 mg (N=6) | Part 1: GSK3640254 200 mg (N=6) | Part 1: Placebo (N=2) | Part 2: GSK3640254 40 mg (N=6) | Part 2: GSK3640254 80 mg (N=6) | Part 2: GSK3640254 140 mg (N=6) | Part 2: Placebo (N=2)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insulin resistance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT03784079/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT03784079/SAP_001.pdf